

Bioequivalence Pivotal Study Protocol of Paroxetine tablets 20 mg under fasting conditions.

### PROJECT NO. / PROTOCOL NO.: AS/BK/OCT-19/0055

Sponsor Code: 212969

#### TITLE

An oral single-dose, randomized, balanced, open-label, two-sequence, two-treatment, two-period, crossover bioequivalence study of Paroxetine tablets 20 mg of GlaxoSmithKline Pharmaceuticals S.A, with that of PAXIL (Paroxetine) tablets 20 mg of GlaxoSmithKline México S.A. de C.V., in healthy adult male and female subjects under fasting conditions.

Version No.: 02

Date: 12/Oct/2020

| CONTRACT RESEARCH ORGANIZATION | SPONSOR |
|---|---|
| Avant Santé Research Center S.A. de C.V. Av. Lázaro Cárdenas No. 500 Col. Residencial San Agustín San Pedro Garza García, Nuevo León México, C.P. 66260 Tel.: PPD www.avantsante.com | GlaxoSmithKline México, S.A. de C.V.<br>Calzada México Xochimilco No. 4900 Col.<br>San Lorenzo Huipulco 14370 Ciudad de<br>México. |

#### **CONFIDENTIALITY STATEMENT**

The information contained and/or attached to this document controlled by the quality system, as well as its formats and/or related registries, is confidential information property of Avant Santé Research Center S.A. de C.V and GlaxoSmithKline México, S.A. de C.V. Any unauthorized use or violation to this notice is prohibited and may be subject to sanctions under applicable law.



Bioequivalence Pivotal Study Protocol of Paroxetine tablets 20 mg under fasting conditions.

### CONTACT INFORMATION OF SPONSOR / INVESTIGATOR

# **Sponsor:**

GlaxoSmithKline México, S.A. de C.V.

Calzada México Xochimilco No. 4900 Col.

San Lorenzo Huipulco 14370 Ciudad de México

# **Primary Study Manager:**

| PPD |
|---------------------------------------------|
| PPD |
| GlaxoSmithKline México, S.A. de C.V. |
| Calzada México Xochimilco No. 4900 Col. |
| San Lorenzo Huipulco 14370 Ciudad de México |
| Phone number: PPD |
| Email: PPD |

# **Sponsor's Authorized Signatory:**

Sigfrido Manuel Rangel Frausto

GlaxoSmithKline México, S.A. de C.V.

Calzada México Xochimilco No. 4900 Col.

San Lorenzo Huipulco 14370 Ciudad de México

Phone number: PPD
Email: PPD

Project No./Protocol No.: AS/BK/OCT-19/0055 Sponsor Code: 212969

Version No: 02 (12/Oct/2020)




Bioequivalence Pivotal Study Protocol of Paroxetine tablets 20 mg under fasting conditions.

# Name and address of Principal Investigator:

Dr. Javier Jesús Osorio Escobar

Avant Santé Research Center S.A. de C.V.

Avenida Lázaro Cárdenas No. 500, Col Residencial San Agustín, San Pedro Garza García, Nuevo

León., México, C.P 66260. Tel.: PPD extension -PPD.

E-mail: PPD

# Name and address of Clinical Investigator:

Dr. José Guillermo Sander Padilla

Avant Santé Research Center S.A. de C.V.

Avenida Lázaro Cárdenas No. 500, Col Residencial San Agustín, San Pedro Garza García, Nuevo

León., México, C.P 66260 Tel.: PPD extension PPD.

E-mail: PPD



Bioequivalence Pivotal Study Protocol of Paroxetine tablets 20 mg under fasting conditions.

**Author:** This protocol is prepared based on the available literature and applicable regulatory requirements to the best of my knowledge, as well as of previous experience from the sponsor GlaxoSmithKline México, S.A. de C.V.

| Name: | Signature and Date: |
|---|---|
| STATEMENT | OF COMPLIANCE |
| We, the undersigned have read and understood t | his protocol and hereby agree to conduct the study in |
| accordance with the same and to comply with | h all the requirements regarding the obligations of |
| investigators and all other pertinent requireme | nts of the NOM 177-SSA1-2013 (COFEPRIS), the |
| Declaration of Helsinki, the ICH Guidelines on | Good Clinical and Laboratory Practices (WHO) of |
| COFEPRIS and all internal relevant SOPs. We f | further agree to ensure that all the personnel involved |
| in the conduct of this study are duly informed re | egarding their obligations. |
| Signature: | Date: |
| Dr. Javier Jesús Osorio Escobar | |
| Principal Investigator | |
| Signature: | Date: |
| Dr. José Guillermo Sander Padilla | |
| Clinical Investigator | |

Project No./Protocol No.: AS/BK/OCT-19/0055  Version No: 02 (12/Oct/2020)


Sponsor Code: 212969



| Signature: Date: | |
|------------------|-------|
| Biol. PPD | |
| PPD | |
| Signature: | Date: |
| PPD , PhD. | |
| PPD | |
| Signature: | Date: |
| PPD , PhD. | |
| PPD | |



Bioequivalence Pivotal Study Protocol of Paroxetine tablets 20 mg under fasting conditions.

# SANITARY RESPONSIBLE AND QUALITY ASSURANCE

| Signature: | | <b>Date:</b> |
|------------|-----------------------------|--------------|
| Q.F.B PPD | | |
| PPD | | |
| | | _ |
| Signature: | | <b>Date:</b> |
| M. Sc. PPD | | |
| PPD | | |
| Signature: | | <b>Date:</b> |
| M.B.A. PPD | | |
| PPD | (Clinical and Bioanalytical | Unit) |



Bioequivalence Pivotal Study Protocol of Paroxetine tablets 20 mg under fasting conditions.

### SPONSOR'S APPROVAL

I, the undersigned, have read and understood this protocol and agree hereby to have the study conducted in accordance with the same and to comply with all the requirements regarding the obligations of Sponsor and all other pertinent requirements of the current NOM-177-SSA1-2013 (COFEPRIS), of the Declaration of Helsinki, ICH Guidelines on Good Clinical and Laboratory Practices (WHO) and of COFEPRIS.

| | Date: |
|-------------------------|-------|
| Authorization Signature | |

# **Sigfrido Manuel Rangel Frausto**

GlaxoSmithKline México, S.A. de C.V.

Calzada México Xochimilco No. 4900 Col.

San Lorenzo Huipulco 14370 Ciudad de México

Ph. No.: PPD

...

Email: PPD




Bioequivalence Pivotal Study Protocol of Paroxetine tablets 20 mg under fasting conditions.

# **TABLE OF CONTENTS**

| TITLE | E 1 | |
|--------|------------------------------------------------------|----|
| CONT | TACT INFORMATION OF SPONSOR / INVESTIGATOR | 2 |
| STAT | EMENT OF COMPLIANCE | 4 |
| SANIT | TARY RESPONSIBLE AND QUALITY ASSURANCE | 6 |
| SPON | SOR'S APPROVAL | 7 |
| TABL | E OF CONTENTS | 8 |
| LIST ( | OF FIGURES | 11 |
| LIST ( | OF TABLES | 11 |
| 1.0 | PROTOCOL SUMMARY | 15 |
| 2.0 | STUDY RELATED SERVICES | 25 |
| 3.0 | BACKGROUND INFORMATION | 26 |
| 3.1 | Mechanism of Action | 27 |
| 3.2 | Therapeutic Indications | 28 |
| 3.3 | Pharmacokinetics | 28 |
| 3.3.1 | Absorption | 28 |
| 3.3.2 | Distribution | 29 |
| 3.3.3 | Metabolism | 29 |
| 3.3.4 | Excretion | 29 |
| 3.4 | Dosage and Administration: | 30 |
| 3.5 | Interactions | 30 |
| 4.0 | STUDY OBJECTIVES | 36 |
| 4.1 | Primary Objective | 36 |
| 4.2 | Secondary Objective | 36 |
| 5.0 | HYPOTHESIS OF THE STUDY | 36 |
| 6.0 | STUDY RATIONALE | 37 |
| 6.1 | Dose Rationale | 38 |
| 7.0 | STUDY DESIGN | 38 |
| 7.1 | Study Design | 38 |
| 7.2 | Rationale for Study Design and Blood Sampling Points | 39 |
| 7.3 | Sample Size | 40 |
| 7.4 | Justification of the Sample Size | 40 |

Project No./Protocol No.: AS/BK/OCT-19/0055

Sponsor Code: 212969




# Bioequivalence Pivotal Study Protocol of Paroxetine tablets 20 mg under fasting conditions.

| 7.5 | Washout Period | 41 |
|------|------------------------------------------------------|----|
| 7.6 | Duration of the Study | 42 |
| 7.7 | Randomization | 42 |
| 7.8 | Blinding | 42 |
| 7.9 | Test and Reference Products | 42 |
| 7.10 | Reception and Storage of Investigational Products | 43 |
| 7.11 | Accounting of Investigational Products | 45 |
| 7.12 | Dispensing | 45 |
| 8.0 | SELECTION AND WITHDRAWL OF SUBJECTS | 46 |
| 8.1 | Screening (selection and enrollment) | 46 |
| 8.2 | Clinical Laboratory Tests | 47 |
| 8.3 | Inclusion Criteria | 48 |
| 8.4 | Exclusion Criteria | 49 |
| 8.5 | Criteria for Subject Withdrawal from the Study | 51 |
| 9.0 | TREATMENT OF SUBJECTS | 53 |
| 9.1 | Drug Administration | 53 |
| 9.2 | Dietary Plan | 53 |
| 9.3 | Restrictions | 54 |
| 9.4 | Housing | 56 |
| 9.5 | Sampling Schedule | 57 |
| 9.6 | Sample Processing and Storage | 59 |
| 9.7 | Sample transfer | 59 |
| 10.0 | ASSESSMENT OF EFFICACY | 60 |
| 11.0 | ASSESSMENT OF SAFETY (CLINICAL SAFETY MEASURES) | 60 |
| 11.1 | Recording of Vital Signs and Medical Examination | 60 |
| 11.2 | Identification, Handling and Reporting of AE and SAE | 61 |
| 12.0 | BIOANALYSIS | 70 |
| 12.1 | Sample analysis | 70 |
| 12.2 | Reporting of drug concentration data | 70 |
| 13.0 | PHARMACOKINETIC PARAMETERS | 71 |
| 14.0 | STATISTICAL ANALYSIS | 72 |


Sponsor Code: 212969




# Bioequivalence Pivotal Study Protocol of Paroxetine tablets 20 mg under fasting conditions.

| 14.1 | Descriptive Statistics | 73 |
|---|---|---|
| 14.2 | Analysis of Variance | 74 |
| 14.3 | Statistical Model | 74 |
| 14.4 | Two One-Sided Test for Bioequivalence | 74 |
| 14.5 | Statistical Power | 75 |
| 14.6 | Ratio Analysis | 75 |
| 14.7 | Intra-Subject Variability | 75 |
| 14.8 | Analysis of Outliers | 75 |
| 14.9 | Criteria for elimination of subject data from the statistical analysis. | 76 |
| 14.10 | Bioequivalence Criteria | 77 |
| 15.0 | AMENDMENTS AND PROTOCOL DEVIATIONS | 77 |
| 16.0 | TERMINATION OF A STUDY | 79 |
| 17.0 | DIRECT ACCESS TO SOURCE DATA/DOCUMENTS | 79 |
| 18.0 | QUALITY CONTROL AND QUALITY ASSURANCE | 81 |
| 19.0 | INVESTIGATOR AND DELEGATION OF DUTIES | 81 |
| 20.0 | ETHICAL CONSIDERATIONS | 81 |
| 20.1 | Ethical Standards | 81 |
| 20.2 | Research Ethics Committee and Research Committee | 82 |
| 20.3 | Informed Consent Process | 82 |
| 20.4 | Subject Participation Compensation | 83 |
| 20.5 | Subject's Insurance | 83 |
| 21.0 | DATA HANDLING AND RECORD KEEPING | 83 |
| 21.1 | Clinical Study Report | 84 |
| 21.2 | Confidentiality of Data | 84 |
| 21.3 | Archiving | 84 |
| 21.4 | Publication Policy | 85 |
| 22.0 | LIST OF ATTACHMENTS | 85 |
| 23.0 | REFERENCES | 86 |



Bioequivalence Pivotal Study Protocol of Paroxetine tablets 20 mg under fasting conditions.

# **LIST OF FIGURES**

| Figure 1 Paroxetine structural formula | 27 |
|------------------------------------------------------------------|----|
| Figure 2 Study Design Diagram | 39 |
| LIST OF TABLES | |
| Table 1 Pharmacokinetic Parameters of Paroxetine | 30 |
| Table 2 Adverse reactions of Paroxetine | 34 |
| Table 3 Investigational Product Details | 42 |
| Table 4 Laboratory Tests | 47 |
| Table 5 Nutritional value of diet on study day 1 | 54 |
| Table 6 Blood volume of samples to be collected during the study | 57 |
| Table 7 Adverse Reaction Classification | 65 |
| Table 8 Pregnancy follow up | 69 |

Project No./Protocol No.: AS/BK/OCT-19/0055  Version No: 02 (12/Oct/2020) Sponsor Code: 212969



#### Bioequivalence Pivotal Study Protocol of Paroxetine tablets 20 mg under fasting conditions.

#### **ABBREVIATIONS**

ADR(s) : Adverse Drug Reaction(s)

AE(s) : Adverse Event(s)
ANOVA : Analysis of Variance

AUC<sub>0-inf</sub> : Area Under Plasma Concentration-Time Curve from Time 0 to Infinite

Area Under Plasma Concentration-Time Curve from Time Zero to the Last Measurable

AUC<sub>0-t</sub> : Concentration

BLOQ : Below the Limit of Quantification

BMI : Body Mass Index

C<sub>max</sub>: Maximum Concentration Observed in Plasma

Federal Commission for the Protection against Sanitary Risk (Comisión Federal para la

Prevención contra Riesgos Sanitarios)

CNFV : Pharmacovigilance National Center (Centro Nacional de Farmacovigilancia)

CNS : Central Nervous System
CoA : Certificate of Analysis
COVID-19 : The coronavirus disease

. The colonavirus disease

COX-2 : Cyclooxygenase-2
CRF(s) : Case Report Form(s)

CV : Coefficient of Variation

CYP : Cytochrome P

ECG : Electrocardiogram

GCP : Good Clinical Practices
GLP : Good Laboratory Practices

H : Hour

HIV : Human Immune Deficiency Virus

ICF : Informed Consent Form

ICH : International Council for Harmonization

ICU : Intensive Care Unit

IP(s) : Investigational Product(s)

Kg : Kilogram


Sponsor Code: 212969




### Bioequivalence Pivotal Study Protocol of Paroxetine tablets 20 mg under fasting conditions.

L Liter

LOQ Limit of quantification

M Missing Sample  $m^2$ Square Meter

**MAOIs** Monoamine Oxidase Inhibitors

Milligram mg mLMilliliter

mmHg Millimeter of Mercury

Nanogram Ng

NOM Mexican Official Norm

**NSAIDs** Nonsteroidal Anti-Inflammatory Drugs

OCD Obsessive Compulsive Disorder

OTC Over-the-counter Potential hydrogen рН PΙ Principal Investigator Quality Assurance QA OC Quality Control OT O-wave and T-wave

REC/RC Research Ethics Committee / Research Committee

**RLS** Restless Legs Syndrome Research Master File **RMF** Rpm Revolutions Per Minute

RT-PCR Real time-Polymerase Chain Reaction Serious Adverse Drug Reaction(s) SADR(s)

SAE(s) Serious Adverse Event(s)

SARS-CoV-2 Severe Acute Respiratory Syndrome Coronavirus 2

SAS Statistical Analysis System

SGPT/ALT Serum Glutamate Pyruvate Transaminase / Alanine Transferase

SGOT/AST Serum Glutamate Oxaloacetate Transaminase / Aspartate Transferase

**SIADH** Syndrome of Inappropriate Anti-Diuretic Hormone Secretion

SOP(s) Standard Operating Procedure

Sponsor Code: 212969




### Bioequivalence Pivotal Study Protocol of Paroxetine tablets 20 mg under fasting conditions.

SSRIs : Selective Serotonin Reuptake Inhibitors

 $t_{1/2}$  : Half-Life

TCAs : Tricyclic Antidepressants
THC : Tetra Hydro Cannabinoids

TMF : Trial Master File

 $T_{max}$  : Time of the Maximum measured plasma concentration

UADR(s) : Unexpected Adverse Drug Reaction(s)

UPLC : Ultra Performance Liquid ChromatographyUSFDA : United States Food and Drug Administration

VDRL : Venereal Disease Research Laboratory

% : Percent

<sup>0</sup>C : Degree Celsius μg : Microgram

5-HT : 5-hydroxytryptamine




Sponsor Code: 212969

Format No.: CPF127-03E No. Reference SOP: CP006

Bioequivalence Pivotal Study Protocol of Paroxetine tablets 20 mg under fasting conditions.

#### 1.0 PROTOCOL SUMMARY

| | An oral single-dose, randomized, balanced, open-label, two-sequence, two- |
|---|---|
| | treatment, two-period, crossover bioequivalence study of Paroxetine tablets 20 mg |
| Study Title | of GlaxoSmithKline Pharmaceuticals S.A, with that of PAXIL (Paroxetine) |
| | tablets 20 mg of GlaxoSmithKline México S.A. de C.V., in healthy adult male |
| | and female subjects under fasting conditions. |
| Regulatory | |
| Agency and | COFEPRIS-México. |
| Country of | COPERNS-MEXICO. |
| Submission | |
| | Primary Objective: |
| | To evaluate and compare the single oral dose bioavailability of Paroxetine tablets |
| | 20 mg manufactured by GlaxoSmithKline Pharmaceuticals S.A. for |
| Study | GlaxoSmithKline México, S.A. de C.V. with that of PAXIL (Paroxetine) tablets |
| <b>Objective</b> | 20 mg of GlaxoSmithKline México, S.A. de C.V. in healthy, adult, male and |
| Objective | female subjects under fasting conditions. |
| | Secondary Objective: |
| | To evaluate safety and tolerability of single oral dose of Paroxetine 20 mg tablets |
| | in healthy adult male and female subjects under fasting conditions. |
| Study Design | An oral single-dose, randomized, balanced, open-label, two-sequence, two- |
| Study Design | treatment, two-period, crossover bioequivalence study under fasting conditions. |
| Sample Size | At least 34 healthy adult male and female subjects will be randomized and dosed |
| Sample Size | in this study. |
| | l |




# Bioequivalence Pivotal Study Protocol of Paroxetine tablets 20 mg under fasting conditions.

| | Test product (A): Paroxetine tablets 20 mg. |
|---|---|
| | [Paroxetine as Paroxetine hydrochloride]. |
| | Manufactured by: GlaxoSmithKline Pharmaceuticals S.A. |
| Study | Manufactured for: GlaxoSmithKline México, S.A. de C.V. |
| Treatments | Reference product (B): PAXIL (Paroxetine as Paroxetine hydrochloride) tablets |
| | 20 mg. |
| | Manufactured by: GlaxoSmithKline México, S.A. de C.V. |
| | Sanitary Registration Number: 008M93SSA IV. |
| | Paroxetine is an antidepressants drug. It is the hydrochloride salt of a |
| | phenylpiperidine compound identified chemically as (-)-trans-4R- |
| | (4'fluorophenyl)-3S-[(3',4'-methylenedioxyphenoxy) methyl] piperidine |
| | hydrochloride hemihydrate and has the empirical formula of |
| | $C_{19}H_{20}FNO_3 \bullet HCl \bullet 1/2H_2O.$ |
| | Paroxetine is indicated for the treatment of: |
| Introduction | Major depressive disorder. |
| | Obsessive Compulsive Disorder (OCD). |
| | Panic disorder with and without agoraphobia. |
| | Social anxiety disorders/social phobia. |
| Generalised anxiety disorder. | |
| | Post-traumatic stress disorder. |
| Screening | Healthy adult male & female volunteers, light or non or ex-smokers, aged between |
| (selection and | 18 and 55 years (both inclusive), with a weight $\geq$ 50.00 kg, with a BMI between $\geq$ 18.0 and $\leq$ 27.0 kg/m <sup>2</sup> will be selected according to the inclusion and exclusion |
| enrollment) | |
| om omnent) | criteria. |


Sponsor Code: 212969



Sponsor Code: 212969

Format No.: CPF127-03E No. Reference SOP: CP006

# Bioequivalence Pivotal Study Protocol of Paroxetine tablets 20 mg under fasting conditions.

| | All the subjects will have a medical history during the selection and enrollment |
|---|---|
| | process. |
| | Volunteers shall be found healthy according to the physical examination |
| | (including vital signs assessment), normal laboratory test results and 12-l |
| | ECG. |
| | The physical examination findings, ECG and laboratory tests will be considered |
| | valid for a maximum period of 90 days prior to the dosing on the first period of |
| | the study. |
| | Pregnancy test in urine will be carried out during the screening period and at the |
| | time of each period check-in for all female subjects. |
| | Real-time (RT-PCR) test for the detection and diagnosis of SARS-COV-2 will be |
| | carried out within the 72 hours prior to the first period check-in for all the subjects. |
| | Avant Santé Research Center S.A. de C.V. will ensure the volunteer participation |
| | history by verifying the COFEPRIS database for bioequivalence studies. |
| | In each study period, all subjects will be required to fast overnight for at least |
| | 10.00 hours prior to dosing until at least 04.00 hours post-dose. |
| | In each study period, a single-dose of either the test product (A) or reference |
| | product (B) will be orally administered to the subjects in sitting posture along with |
| | 250 mL of water at room temperature under fasting conditions. |
| Drug | The administration of the test or reference products to each subject will be |
| Administration | performed as per a randomization schedule. |
| (Dosing) | The subjects will be instructed to swallow the tablet as a whole as mentioned in |
| | the prescribing information and not to touch the tablet with their hands, chew or |
| | crush the tablet since this can affect the drug release. |




# Bioequivalence Pivotal Study Protocol of Paroxetine tablets 20 mg under fasting conditions.

| | Hands and mouth will be checked after dosing to ensure compliance and a |
|---|---|
| | subject does not touch the IP with hands. |
| | Immediately after dosing in each period trained study personnel will evaluate the |
| | compliance by supervising the complete administration procedure SOP CP020 |
| | (Administration of the Investigational Product). |
| | Drug administration will be registered in the respective source documents. |
| | Subjects will be provided with standard meals throughout their stay in the |
| | facilities. |
| | On the check-in day (day -1) they will receive dinner, which will be finished at |
| | the latest 10.00 hours prior to dosing at the following day in each study period. |
| D' ( DI | Subjects will be required to fast overnight for at least 10.00 hours prior to dosing |
| Dietary Plan | and until at least 04.00 hours post-dose in each study period. |
| | After the dose administration of test or reference product (day 1), lunch, snack |
| | and dinner will be provided at 04.00, 08.00 and 12.00 (with a grace period of + 45 |
| | minutes) hours post-dose respectively, in each study period. |
| | The meal plan will be uniform for all the subjects and same between the study |
| | periods. |
| | Information on the amount of meal consumed and the time of consumption by |
| | each subject will be registered in the respective source documents. |
| | All subjects will be instructed to follow the below mentioned restrictions for at |
| | least 72.00 hours prior to dosing and till last blood sample collection in each study |
| Study | period: |
| Restrictions | Smoking of cigarettes or nicotine containing products. |
| | • Any food or beverages containing xanthine- (tea, coffee, theobromine, |
| | theophylline, chocolates, cola drinks, etc.). |

Project No./Protocol No.: AS/BK/OCT-19/0055  Version No: 02 (12/Oct/2020) Sponsor Code: 212969




Bioequivalence Pivotal Study Protocol of Paroxetine tablets 20 mg under fasting conditions.

Alcohol or related products.

Smoked or carbon cooked food.

Beverages with pomelos or grapefruit juice or products containing

grapefruit extract (e.g. soda).

Medications

All subjects will be asked about their medication history. They will be instructed not to take any medication until the study is completed; particularly during the last 14 days preceding the first dosing for any prescribed medication, the last 7 days before for OTC medicinal or herbal products used for therapeutic purposes, and the last 30 days before for any enzyme inhibiting / inducing drugs preceding

the first dosing.

Subjects will be specifically reminded that the restriction mentioned above

includes analgesics, cold & anti-allergic preparations, vitamins and natural

products used for therapeutic benefits and antacid preparations.

Vitamins used as nutritional supplements in non-therapeutic doses (as judged by

the principal investigator or designee) may be accepted, but their consumption

must be stopped from at least 7 days prior to the dosing and until the study is

completed.

Fluid (water) restriction

The subjects will not be allowed to drink water 1 hour before and until 2 hours

post-dose except for the 250 mL of water provided for the dosing, unless it is

clinically indicated; at all other times water will be provided *ad libitum*.

Postural (activity) Restriction

The dose will be administered to all subjects at the scheduled time and subjects

will be instructed to remain in comfortable sitting position for the first 02.00




# Bioequivalence Pivotal Study Protocol of Paroxetine tablets 20 mg under fasting conditions.

| | hours following the drug administration except when clinically indicated or |
|---|---|
| | protocol specified activity (blood sample collection) or due to natural exigencies |
| | After 02.00 hours post-dose, subjects will be allowed to wander and will be |
| | advised to avoid any severe physical exertion. |
| | In case of an adverse event (AE), subjects will be maintained in the proper position |
| | as per physician's assessment in each study period. |
| | Subjects will be in the clinical facility from at least 10.50 hours prior to the dosing |
| | until the last in-house blood sample collection i.e. 24 hours in each study period. |
| | Subjects will visit clinical facility at 36.00, 48.00 and 72.00 hours for the |
| Housing | collection of the ambulatory samples in each study period. |
| | Subjects will be instructed to self-quarantine during the outpatient period of the study i.e. until 72 h blood sample collection in period-2 or until withdrawal, |
| | whichever is earlier, and to monitor at home their daily body temperature. |
| Washout | There will be a washout period of at least 7 days between successive dosing. |
| Period | There will be a washout period of at least / days between successive dosing. |
| | In each study period, a total of 24 blood samples (4 mL each) will be collected |
| | from each subject as per the following schedule: |
| | • The first blood sample will be collected within 1.50 hours prior to the |
| Sampling | dosing (00.00 hours / pre-dose). |
| Schedule | • The remaining samples will be collected after the dosing of the test or |
| | reference drug at 00.50, 01.00, 01.50, 02.00, 02.50, 03.00, 03.50, 04.00, |
| | 04.50, 05.00, 05.50, 06.00, 06.50, 07.00, 08.00, 09.00, 10.00, 12.00, 16.00, |
| | 24.00, 36.00, 48.00 and 72.00 hours. |
| L | , 1 |

Project No./Protocol No.: AS/BK/OCT-19/0055  Version No: 02 (12/Oct/2020) Sponsor Code: 212969



Sponsor Code: 212969

Format No.: CPF127-03E No. Reference SOP: CP006

# Bioequivalence Pivotal Study Protocol of Paroxetine tablets 20 mg under fasting conditions.

| • The samples corresponding to 36.00, 48.00 and 72.00 hours possible collected on separate visits as ambulatory sample in each p | ost dose will |
|---|---|
| he collected on senarate visits as ambulatory sample in each n | |
| be confected on separate visits as amountainly sample in each p | eriod of the |
| study. | |
| The total blood volume collected from each subject will not exceed | ed 223 mL, |
| which includes about 10 mL for the selection process (selection and e | enrollment), |
| 21 mL for the discarded heparinized blood and 192 mL for the pharm | macokinetic |
| evaluation. | evaluation. |
| If circumstances arise, where more than 223 + 10 mL of blood from | each subject |
| needs to be withdrawn the subject will be asked for additional conser | nt and REC / |
| RC will be informed. | |
| Once collected, the blood samples will be placed in an ice-filled | container or |
| another cooling device until the centrifugation process is started. | |
| Centrifugation process will be started within 45 minutes from the ti | me of blood |
| sample collection and will be performed at 3000 rpm for 10 minutes | at $4 \pm 2$ °C. |
| Blood Sample The plasma obtained from blood samples will be transferred as soon | ı as possible |
| Collection, into two different cryo-tubes (aliquot 1 and aliquot 2), pre-labeled | with project |
| Processing and number, period number, subject number, sample number and aliquot | number. |
| Storage The plasma volume obtained from blood sample will be allocated as | follows: |
| Aliquot 1: 1.0 mL of plasma (approximately). | |
| Aliquot 2: rest of the plasma. | |
| All plasma samples (aliquot 1 for sample analysis and aliquot 2 as b | ack-up) will |
| be stored at a temperature of -50 °C or below. | |
| Safety Medical examination will be performed before check-in, prior to the | e dosing and |
| <b>Assessment</b> before the check-out in each study period. | |




#### Bioequivalence Pivotal Study Protocol of Paroxetine tablets 20 mg under fasting conditions.

Nevertheless, it may also be performed at any time during the study conduction if judged necessary by the physician.

Physical examination will be performed before check-in of each study period and

Physical examination will be performed before check-in of each study period and may also be performed at any time during the study conduction if judged necessary by the physician.

Vital signs (sitting blood pressure, pulse rate, respiratory rate and axillary-body temperature) will be measured and registered at the time of check-in, prior to dosing, at 03.00, 05.00 and 12.00 hours (within  $\pm 45$  minutes) after the dosing, before the check-out and at the time of each ambulatory sample collection in each study period.

The subjects' well-being will be asked at the time of the medical examination, during the vital signs recording and at the time of each ambulatory sample collection in each study period; this will be registered in the respective source document.

Seven (7) to 9 days after the collection of 72-h blood sample in second period or after the withdrawal, a telephone call will be made to each subject by the personnel designated by the PI to monitor any serious adverse event, specifically, subjects will be questioned about any symptoms related to COVID-19.

# Bioanalysis

Sponsor Code: 212969

The concentration of Paroxetine in plasma samples collected during the study will be quantified using a validated bioanalytical UPLC/MS-MS method (LOQ - 0.106 ng/mL) according to COFEPRIS guidelines, GLP and in-house SOPs.

Method validation and subject sample analysis will be performed using same anticoagulant (K<sub>2</sub>-EDTA) that will be used for blood sample collection in clinical phase.




# Bioequivalence Pivotal Study Protocol of Paroxetine tablets 20 mg under fasting conditions.

| | Employing the observed concentration vs. time profiles of Paroxetine and using |
|---|---|
| Pharmacokinetic Parameters | WinNonlin® software (version 6.4 or higher), the following pharmacokinetic |
| | parameters will be calculated: |
| | <ul> <li>Primary Variables: C<sub>max</sub> and AUC<sub>0-t.</sub></li> </ul> |
| | • Secondary Variables: AUC <sub>0-inf</sub> , AUC_% Extrap, T <sub>max</sub> , Kel, t <sub>1/2</sub> . |
| | Descriptive statistics will be calculated. Statistical analysis will be performed by |
| Statistical | using ANOVA on ln-transformed pharmacokinetic parameters $C_{\text{max}}$ and $AUC_{0\text{-t.}}$ |
| Analysis | The statistical model used in this research is a general linear model and the same |
| | is covered in protocol section 14.3 |
| | Based on the statistical results of classic 90% confidence interval for the ratio of |
| | the geometric least squares means for In-transformed pharmacokinetic |
| | parameters $C_{\text{max}}$ and $AUC_{0\text{-t}}$ for Paroxetine conclusion will be drawn for test |
| | product (A) vs. the reference product (B) under fasting conditions. |
| BE Criteria | The bioequivalence of the test product (A) with that of the reference product (B) |
| DE CITCHA | under fasting conditions will be concluded, if the 90% Confidence Intervals of the |
| | ratio of the test and reference product (test/reference) falls within the acceptance |
| | range of $80.00-125.00\%$ for the In-transformed parameters $C_{\text{max}}$ and $AUC_{0\text{-t}}$ for |
| | Paroxetine. |
| | This study will be conducted carried as per NOM-177-SSA1-2013, COFEPRIS |
| Ethical | guidelines, ICH-GCP and principles of Declaration of Helsinki (Fortaleza, Brazil, |
| | October 2013). |
| Considerations | Protocol, Case Report Form (CRF) and the informed consent form (ICF) approval |
| | will be taken from the REC / RC, and COFEPRIS before initiation of the study. |

Project No./Protocol No.: AS/BK/OCT-19/0055  Version No: 02 (12/Oct/2020) Sponsor Code: 212969

Avant Santé Research Center S.A. de C.V



# Bioequivalence Pivotal Study Protocol of Paroxetine tablets 20 mg under fasting conditions.

| Clinical Study<br>Report | The clinical study report will be prepared as per NOM-177-SSA1-2013 (COFEPRIS) and sponsor requirements, having all the clinical, bioanalytical, pharmacokinetic and statistical data subjected to Quality Assurance audits. |
|---|---|
| Archiving | The raw data and reports will be filed at Avant Santé Research Center S.A. de C.V, with controlled access for 30 years. Avant Santé Research Center S.A. de C.V. will not destroy/discard any document related to the study without written confirmation from the sponsor. |




Bioequivalence Pivotal Study Protocol of Paroxetine tablets 20 mg under fasting conditions.

### 2.0 STUDY RELATED SERVICES

#### 2.1 Research Ethics Committee

Research Ethics Committee of Avant Santé Research Center S.A. de C.V.,

Av. Lázaro Cárdenas # 500, Col. Residencial San Agustín,

San Pedro Garza García, N. L.,

México, C. P. 66260.Tel: PPD to PPD

#### 2.2 Research Committee

Research Committee of Avant Santé Research Center S.A. de C.V.,

Av. Lázaro Cárdenas # 500, Col. Residencial San Agustín,

San Pedro Garza García, N. L.,

México, C. P. 66260.Tel: PPD to PPD.

### 2.3 Clinical Diagnostic Laboratory

• Swiss Lab (SwissLab S.A. de C.V.)

Río San Juan 200, Miravalle, CP 64660.

Monterrey, N.L. México, Tel. PPD

and / or

• Grupo Diagnóstico Médico Proa S.A. de C.V. (This lab is considered as a back-up)

Alfonso Herrera 75, Col. San Rafael, Delegación Cuauhtémoc. Ciudad de México.

México. CP 06470. Tel: PPD

# 2.4 Contract Hospital

Swiss Hospital S.A.P.I. de C.V.,

Río San Juan # 200, Colonia Miravalle, Monterrey, Nuevo León, México,

C.P. 64650, Tel: PPD , Emergencies: PPD

#### 2.5 Ambulance

Sponsor Code: 212969




### Bioequivalence Pivotal Study Protocol of Paroxetine tablets 20 mg under fasting conditions.

Emergencia Médica Profesional, S. C.

Calzada San Pedro No. 504-A, Colonia Fuentes del Valle, San Pedro Garza García, Nuevo

León. C.P. 66220

Tel: PPD , Emergency: PPD

#### 2.6 Clinical Unit

Avant Santé Research Center S.A. de C.V.

Ave. Lázaro Cárdenas No. 500, Col. Residencial San Agustín, San Pedro Garza García,

Nuevo León, México, C.P. 66260

Tel.: PPD to PPD

### 2.7 Bioanalytical Unit

Avant Santé Research Center S.A. de C.V.

Ave. Lázaro Cárdenas No. 500,

Col. Residencial San Agustín, San Pedro Garza García, Nuevo León, México, C.P. 66260

Tel.: PPD to PPD

#### 2.8 Biostatistics Service

Avant Santé Research Center S.A. de C.V.

Ave. Lázaro Cárdenas No. 500, Col. Residencial San Agustín,

San Pedro Garza García, Nuevo León, México, C.P. 66260

Tel.: PPD to PPD

#### 2.9 Biological Waste Management

Veolia Soluciones Industriales México, S.A de C.V

Av. Lázaro Cárdenas No. 435, PISO 10, Col. Zona Loma Larga Oriente

San Pedro Garza García, Nuevo León C.P 66266

Tel.: PPD Fax PPD

e-mail: PPD www.veolia.com.mx

#### 3.0 BACKGROUND INFORMATION

Sponsor Code: 212969




#### Bioequivalence Pivotal Study Protocol of Paroxetine tablets 20 mg under fasting conditions.

Paroxetine is an antidepressant drug <sup>[1]</sup>. It is the hydrochloride salt of a phenylpiperidine compound identified chemically as (-)-trans-4R-(4'fluorophenyl)-3S- [(3',4' methylene di oxy phenoxy) methyl] piperidine hydrochloride hemihydrate and has the empirical formula of  $C_{19}H_{20}FNO_3 \cdot HCl \cdot 1/2H_2O$ . Its molecular weight is 374.8 g/mol. and its structural formula is: <sup>[2]</sup>

Figure 1 Paroxetine hydrochloride structural formula

#### 3.1 Mechanism of Action

Sponsor Code: 212969

Paroxetine is a potent and selective inhibitor of 5-hydroxytryptamine (5-HT, serotonin) reuptake and is thought to be related to its specific inhibition of 5-HT reuptake in brain neurons.

Paroxetine is chemically unrelated to the tricyclic, tetracyclic and other available antidepressants.

Paroxetine has low affinity for muscarinic cholinergic receptors and animal studies have indicated only weak anticholinergic properties.

In accordance with this selective action, *in vitro* studies have indicated that, in contrast to tricyclic antidepressants, paroxetine has little affinity for alpha1, alpha2 and beta-adrenoceptors, dopamine (D2), 5-HT1 like, 5-HT2 and histamine (H1) receptors. This lack




Bioequivalence Pivotal Study Protocol of Paroxetine tablets 20 mg under fasting conditions.

of interaction with post-synaptic receptors in vitro is substantiated by in vivo studies which

demonstrate lack of CNS depressant and hypotensive properties. [1]

**Therapeutic Indications** 3.2

Paroxetine is indicated for the treatment of:

Major depressive disorder.

• Obsessive Compulsive Disorder (OCD).

Panic disorder with and without agoraphobia.

Social anxiety disorders/social phobia.

Generalised anxiety disorder.

Post-traumatic stress disorder. [1]

3.3 Pharmacokinetics

3.3.1 Absorption

Paroxetine is well absorbed after oral dosing and undergoes first-pass metabolism. Due to

first-pass metabolism, the amount of paroxetine available to the systemic circulation is less

than that absorbed from the gastrointestinal tract. Partial saturation of the first-pass effect and

reduced plasma clearance occur as the body burden increases with higher single doses or on

multiple dosing. This results in disproportionate increases in plasma concentrations of

paroxetine and hence pharmacokinetic parameters are not constant, resulting in non-linear

kinetics. However, the non-linearity is generally small and is confined to those subjects who

achieve low plasma levels at low doses.

Steady state systemic levels are attained by 7 to 14 days after starting treatment with

immediate or controlled release formulations and pharmacokinetics do not appear to change

during long-term therapy. [1]


Sponsor Code: 212969




Bioequivalence Pivotal Study Protocol of Paroxetine tablets 20 mg under fasting conditions.

3.3.2 Distribution

Paroxetine is extensively distributed into tissues and pharmacokinetic calculations indicate

that only 1% of the paroxetine in the body resides in the plasma. Approximately 95% of the

paroxetine present is protein bound at therapeutic concentrations.

No correlation has been found between paroxetine plasma concentrations and clinical effect

(adverse experiences and efficacy). [1]

3.3.3 Metabolism

The principal metabolites of paroxetine are polar and conjugated products of oxidation and

methylation which are readily cleared. In view of their relative lack of pharmacological

activity, it is most unlikely that they contribute to paroxetine's therapeutic effects.

Metabolism does not compromise paroxetine's selective action on neuronal 5-HT uptake. [1]

3.3.4 Excretion

Urinary excretion of unchanged paroxetine is generally less than 2% of dose whilst that of

metabolites is about 64% of dose. About 36% of the dose is excreted in faeces, probably via

the bile, of which unchanged paroxetine represents less than 1% of the dose. Thus, paroxetine

is eliminated almost entirely by metabolism.

Metabolite excretion is biphasic, being initially a result of first-pass metabolism and

subsequently controlled by systemic elimination of paroxetine.

[1]

Sponsor Code: 212969




Bioequivalence Pivotal Study Protocol of Paroxetine tablets 20 mg under fasting conditions.

**Table 1 Pharmacokinetic Parameters of Paroxetine** 

| Reference | Drug | Dose<br>(mg) | C <sub>max</sub> (ng/mL) | T <sub>max</sub> (h) | T <sub>1/2</sub> (h) |
|---|---|---|---|---|---|
| 3 (In-house data (Avant Santé) AS/AO/ABR-17/0012 | Paroxetine tablets | 20 mg | 6.884 | 4.806 | 11.4 |
| 4 | Paroxetine tablets | 20 mg | 5.396<br>(µg/L) | 5.35 | 11.98 |

### **Special Populations:**

**Elderly:** Increased plasma concentrations of paroxetine occur in elderly subjects. [1]

# 3.4 Dosage and Administration:

The recommended initial dose is 20 mg daily.

**Administration:** Paroxetine tablets can be administered with or without food. <sup>[2]</sup>

#### 3.5 Interactions

Sponsor Code: 212969

# Interaction with other medicinal products and other forms of interaction:

#### **Serotonergic drugs:**

As with other SSRIs, co-administration with serotonergic drugs may lead to an incidence of 5-HT associated effects. Caution should be advised and a closer clinical monitoring is required when serotonergic drugs (such as L-tryptophan, triptans, tramadol, linezolid, methyl thioninium chloride (methylene blue)), SSRIs, lithium, pethidine and St. John's Wort - Hypericum perforatum - preparations) are combined with paroxetine. Caution is also advised with fentanyl used in general anesthesia or in the treatment of chronic pain.




Bioequivalence Pivotal Study Protocol of Paroxetine tablets 20 mg under fasting conditions.

Concomitant use of paroxetine and MAOIs is contraindicated because of the risk of serotonin

syndrome.

**Pimozide** 

Increased pimozide levels of on average 2.5 times have been demonstrated in a study of a

single low dose pimozide (2 mg) when co-administered with 60 mg paroxetine. This may be

explained by the known CYP2D6 inhibitory properties of paroxetine. Due to the narrow

therapeutic index of pimozide and its known ability to prolong QT interval, concomitant use

of pimozide and paroxetine is contraindicated.

**Drug metabolizing enzymes** 

The metabolism and pharmacokinetics of paroxetine may be affected by the induction or

inhibition of drug metabolizing enzymes.

When paroxetine is to be co-administered with a known drug metabolizing enzyme inhibitor,

consideration should be given to using paroxetine doses at the lower end of the range.

No initial dosage adjustment is considered necessary when the drug is to be co-administered

with known drug metabolizing enzyme inducers (e.g. carbamazepine, rifampicin,

phenobarbital, phenytoin) or with fosamprenavir/ritonavir. Any paroxetine dosage

adjustment (either after initiation or following discontinuation of an enzyme inducer) should

be guided by clinical effect (tolerability and efficacy).

**Neuromuscular Blockers:** 

SSRIs may reduce plasma cholinesterase activity resulting in a prolongation of the

neuromuscular blocking action of mivacurium and suxamethonium.

Fosamprenavir/ritonavir:

Co-administration of fosamprenavir/ritonavir 700/100 mg twice daily with paroxetine 20 mg

daily in healthy volunteers for 10 days significantly decreased plasma levels of paroxetine by

approximately 55%. The plasma levels of fosamprenavir/ritonavir during co-administration

of paroxetine were similar to reference values of other studies, indicating that paroxetine had




Bioequivalence Pivotal Study Protocol of Paroxetine tablets 20 mg under fasting conditions.

no significant effect on metabolism of fosamprenavir/ritonavir. There are no data available

about the effects of long-term co-administration of paroxetine and fosamprenavir/ritonavir

exceeding 10 days.

**Procyclidine:** Daily administration of paroxetine increases significantly the plasma levels of

procyclidine. If anti-cholinergic effects are seen, the dose of procyclidine should be reduced.

Anticonvulsants: carbamazepine, phenytoin, sodium valproate. Concomitant administration

does not seem to show any effect on pharmacokinetic/dynamic profile in epileptic patients.

CYP2D6 inhibitory potency of paroxetine:

As with other antidepressants, including other SSRIs, paroxetine inhibits the hepatic

cytochrome P450 enzyme CYP2D6. Inhibition of CYP2D6 may lead to increased plasma

concentrations of co-administered drugs metabolised by this enzyme. These include certain

tricyclic antidepressants (e.g. clomipramine, nortriptyline, and desipramine), phenothiazine

neuroleptics (e.g. perphenazine and thioridazine), risperidone, atomoxetine, certain Type 1c

antiarrhythmics (e.g. propafenone and flecainide) and metoprolol. It is not recommended to

use paroxetine in combination with metoprolol when given in cardiac insufficiency, because

of the narrow therapeutic index of metoprolol in this indication.

Pharmacokinetic interaction between CYP2D6 inhibitors and tamoxifen, showing a 65-75%

reduction in plasma levels of one of the more active forms of tamoxifen, i.e. endoxifen, has

been reported in the literature. Reduced efficacy of tamoxifen has been reported with

concomitant usage of some SSRI antidepressants in some studies. As a reduced effect of

tamoxifen cannot be excluded, co-administration with potent CYP2D6 inhibitors (including

paroxetine) should whenever possible be avoided.

Alcohol:

As with other psychotropic drugs patients should be advised to avoid alcohol use while taking

paroxetine.


Sponsor Code: 212969




Bioequivalence Pivotal Study Protocol of Paroxetine tablets 20 mg under fasting conditions.

Oral anticoagulants:

A pharmacodynamic interaction between paroxetine and oral anticoagulants may occur.

Concomitant use of paroxetine and oral anticoagulants can lead to an increased anticoagulant

activity and haemorrhagic risk. Therefore, paroxetine should be used with caution in patients

who are treated with oral anticoagulants.

NSAIDs and acetylsalicylic acid, and other antiplatelet agents:

A pharmacodynamic interaction between paroxetine and NSAIDs/acetylsalicylic acid may

occur. Concomitant use of paroxetine and NSAIDs/acetylsalicylic acid can lead to an

increased haemorrhagic risk.

Caution is advised in patients taking SSRIs, concomitantly with oral anticoagulants, drugs

known to affect platelet function or increase risk of bleeding (e.g. atypical antipsychotics such

as clozapine, phenothiazines, most TCAs, acetylsalicylic acid, NSAIDs, COX-2 inhibitors)

as well as in patients with a history of bleeding disorders or conditions that may predispose

to bleeding.

**Pravastatin:** 

An interaction between paroxetine and pravastatin has been observed in studies suggesting

that co-administration of paroxetine and pravastatin may lead to an increase in blood glucose

levels. Patients with diabetes mellitus receiving both paroxetine and pravastatin may require

dosage adjustment of oral hypoglycaemic agents and/or insulin.

Drugs affecting gastric pH:

In vitro data have shown that dissociation of paroxetine from the oral suspension is pH-

dependant. Therefore, drugs that alter gastric pH (such as antacid drugs, proton pump

inhibitors or histamine H2-receptor antagonists) may affect plasma paroxetine concentrations

in patients taking the oral suspension. [1]


Sponsor Code: 212969




Bioequivalence Pivotal Study Protocol of Paroxetine tablets 20 mg under fasting conditions.

### 3.6 Adverse Drug Reactions

Some of the adverse drug reactions listed below may decrease in intensity and frequency with continued treatment and do not generally lead to cessation of therapy. Adverse drug reactions are listed below by system organ class and frequency. Frequencies are defined as: very common ( $\geq 1/10$ ), common ( $\geq 1/100$ ), very rare (<1/1000), uncommon ( $\geq 1/1000$ ), rare ( $\geq 1/10000$ ), very rare (<1/10000), including isolated reports. [1]

**Table 2 Adverse reactions of Paroxetine** 

| System organ class | Frequency | Adverse Reaction |
|---|---|---|
| Blood and lymphatic | Uncommon | Abnormal bleeding, predominantly of the skin and mucous membranes |
| disorders | | (including ecchymosis and gynecological bleeding). |
| | Very rare | Thrombocytopenia. |
| Immune system disorders | Very rare | Severe and potentially fatal allergic reactions (including anaphylactoid reactions and angioedema). |
| Endocrine disorders | Very rare | Syndrome of inappropriate anti-diuretic hormone secretion (SIADH). |
| Metabolism and nutrition | Common | Increases in cholesterol levels, decreased appetite. |
| disorders | Uncommon | Altered glycaemic control has been reported in diabetic patients. |
| | Rare | Hyponatraemia. |
| Psychiatric disorders | Common | Somnolence, insomnia, agitation, abnormal dreams (including |
| | | nightmares). |
| | Uncommon | Confusion, hallucinations. |
| | Rare | Manic reactions, anxiety, depersonalization, panic attacks, akathisia. |
| Nervous system disorders | Common | Dizziness, tremor, headache, concentration impaired. |
| | Uncommon | Extrapiramidal disorders. |
| | Rare | Convulsions, restless legs syndrome (RLS). |
| | Very rare | Serotonin syndrome (symptoms may include agitation, confusion, |
| | | diaphoresis, hallucinations, hyperreflexia, myoclonus, shivering, |
| | | tachycardia and tremor). |
| Eye disorders | Common | Blurred vision. |
| | Uncommon | Mydriasis. |
| | Very rare | Acute glaucoma. |
| Cardiac disorders | Uncommon | Sinus tachycardia. |
| | Rare | Bradycardia. |


Sponsor Code: 212969




### Bioequivalence Pivotal Study Protocol of Paroxetine tablets 20 mg under fasting conditions.

| System organ class | Frequency | Adverse Reaction |
|---|---|---|
| Vascular disorders | Uncommon | Transient increases or decreases in blood pressure, postural hypotension. |
| Respiratory, thoracic and mediastinal disorders | | Yawning. |
| Gastrointestinal disorders | Very common | Nausea. |
| | Common | Constipation, diarrhoea, vomiting and dry mouth. |
| | Very rare | Gastrointestinal bleeding. |
| | Rare | Elevation of hepatic enzymes. |
| Hepatobiliary disorders | Very rare | Hepatic events (such as hepatitis, sometimes associated with jaundice and/or liver failure). |
| | Common | Sweating. |
| Skin and subcutaneous | Uncommon | Skin rashes, pruritus. |
| tissue disorders | Very rare | Severe cutaneous adverse reactions (including erythema multiforme, Stevens-Johnson syndrome and toxic epidermal necrolysis), urticaria, photosensitivity reactions. |
| Renal and urinary disorders | Uncommon | Urinary retention, urinary incontinence. |
| | Very<br>common | Sexual dysfunction. |
| Reproductive system and breast disorders | Rare | Hyperprolactinaemia/galactorrhoea, menstrual disorders (including menorrhagia, metrorrhagia, amenorrhoea, menstruation delayed and menstruation irregular). |
| | Very rare | Priapism. |
| Musculoskeletal and connective tissue disorders Rare | | Arthralgia, myalgia. |
| General disorders and | Common | Asthenia, body weight gain. |
| administration site conditions | Very rare | Peripheral oedema. |

### 3.7 Contraindications

Sponsor Code: 212969

# Paroxetine is contraindicated with following:

- Hypersensitivity to the active substance or to any of the excipients.
- In combination with monoamine oxidase inhibitors (MAOIs including linezolid and methylene blue).




Bioequivalence Pivotal Study Protocol of Paroxetine tablets 20 mg under fasting conditions.

Paroxetine should not be used in combination with thioridazine, because, as with other

drugs which inhibit the hepatic enzyme CYP450 2D6, paroxetine can elevate plasma

levels of thioridazine. Administration of thioridazine alone can lead to QTc interval

prolongation with associated serious ventricular arrhythmia such as torsade's de

pointes, and sudden death.

Paroxetine should not be used in combination with pimozide. [1]

4.0 STUDY OBJECTIVES

4.1 Primary Objective

To evaluate and compare the single oral dose bioavailability of Paroxetine tablets 20 mg

manufactured by GlaxoSmithKline Pharmaceuticals S.A. for GlaxoSmithKline México, S.A.

de C.V. with that of PAXIL (Paroxetine) tablets 20 mg of GlaxoSmithKline México, S.A. de

C.V. in healthy, adult, male and female subjects under fasting conditions.

4.2 Secondary Objective

To evaluate the safety and tolerability of single oral dose of Paroxetine 20 mg tablets in

healthy adult male and female subjects under fasting conditions.

5.0 HYPOTHESIS OF THE STUDY

Null hypothesis: H<sub>0</sub>: mean test / mean reference < L or mean test / mean reference > U

Paroxetine tablets 20 mg manufactured by GlaxoSmithKline Pharmaceuticals S.A. and

PAXIL (Paroxetine) tablets 20 mg of GlaxoSmithKline México, S.A de C.V. are not

bioequivalent.

Alternative hypothesis:  $H_1$ :  $L \le mean test / mean reference \le U$ 

Paroxetine tablets 20 mg manufactured by GlaxoSmithKline Pharmaceuticals S.A. and

PAXIL (Paroxetine) tablets 20 mg of GlaxoSmithKline México, S.A. de C.V. are

bioequivalent.


Sponsor Code: 212969




Bioequivalence Pivotal Study Protocol of Paroxetine tablets 20 mg under fasting conditions.

Two one-sided t-tests will be carried out on each PK parameter of Paroxetine using least

squares means (LSM) values for geometric LSMs of the primary PK parameters (mean test

or mean reference = LSM value of the corresponding PK parameter for test or reference

product). The type I error will be set to  $\alpha = 5\%$  and therefore 90% (two-tailed) confidence

intervals will be provided together with the indication whether the null hypothesis of

nonequivalence for the appropriate parameter can be rejected.

Probabilities p(t) of Schuirmann, left tail  $(t_l)$  and right tail  $(t_r)$  values will be calculated for the

lower limit L = 0.80 and upper limit +U = 1 / 0.80 = 1.25 for geometric LSM of

pharmacokinetic parameters C<sub>max</sub> and AUC<sub>0-t</sub>.

6.0 STUDY RATIONALE

Paxil (Paroxetine) tablets 20 mg of GlaxoSmithKline México, S.A. de C.V. is listed as a

reference product by COFEPRIS. Currently, the drug product is manufactured at Xochimilco,

México site using wet granulation process and Xochimilco, México site will exit GSK

network in 2021.

Considering the same, Paroxetine tablets 20 mg manufactured using direct compression

process at GlaxoSmithKline Pharmaceuticals S.A. site was selected as new supplier.

Additionally, formulation composition is modified with respect to in-active ingredients.

To register the above mentioned changes [change in the drug product manufacturing site,

differences in the formulations and process] in the marketing registration application for

México, a bioequivalence study is required as per Oficio Circular CAS/OR/01/868/2013 <sup>[5]</sup> to

establish similarity between the test product (new) manufactured at GlaxoSmithKline

Pharmaceuticals S.A. and reference product manufactured at Xochimilco, México site.

México.




Bioequivalence Pivotal Study Protocol of Paroxetine tablets 20 mg under fasting conditions.

This product is an immediate release product and can be administered with or without food;

hence, the test product (to be marketed) should be bioequivalent to the reference product

under fasting conditions determined by C<sub>max</sub> and AUC<sub>0-t</sub> values of Paroxetine

Hence, the test product PAXIL (Paroxetine) tablets 20 mg manufactured by GlaxoSmithKline

Pharmaceuticals S.A. manufactured for GlaxoSmithKline México S.A. de C.V. will be

compared with that of Paxil (Paroxetine) tablets 20 mg GlaxoSmithKline México, S.A. de

C.V. to evaluate bioequivalence.

6.1 Dose Rationale

The recommended initial dose of Paroxetine is 20 mg/day. Hence, 20 mg dose of Paroxetine

is within the dose range, which is expected to be tolerable in healthy adult volunteers. [2]

7.0 STUDY DESIGN

Each period will have identical procedures. For a detailed schedule of events, see Attachment-

II.

7.1 Study Design

An oral single-dose, randomized, balanced, open-label, two-sequence, two-treatment, two-

period, crossover bioequivalence study under fasting conditions.

The study design is presented in Figure 2 below.


Sponsor Code: 212969 Version No. 02 (12/06/2020)




Bioequivalence Pivotal Study Protocol of Paroxetine tablets 20 mg under fasting conditions.



Figure 2 Study Design Diagram

# **Rationale for Study Design and Blood Sampling Points**

Generally, bioequivalence studies are conducted in healthy adult volunteers. As this product is indicated for men and women, this bioequivalence study is planned in healthy adult human male and female volunteers. These products are an immediate release formulation and it can be administered with or without food, fasting bioequivalence study is required.

In this study two formulations are being compared, a randomised, two-period, two-sequence single dose crossover fasting study design is planned in healthy subjects to assess bioequivalence.

Sampling points have been placed with sufficient frequency to characterize  $C_{max}$  and AUC parameters adequately, considering the  $T_{max}$  and half-life of Paroxetine. The  $T_{max}$  occurs approximately 5.00 hours after the drug administration and the mean elimination half-life is approximately 12 hours [3].

A minimum of seven times the mean half-life will be considered as wash-out period between consecutive treatments to avoid carry-over effects, hence a wash-out period of at least 7 days




Bioequivalence Pivotal Study Protocol of Paroxetine tablets 20 mg under fasting conditions.

is considered. The duration of blood sampling is planned till 72.00 hours to cover at-least four

half-lives for Paroxetine.

7.3 Sample Size

At least 34 healthy adult male and female subjects are required to meet at least a statistical

power of 90% at 5% level of significance to achieve the bioequivalence results within 80.00-

125.00% in this study. In addition, a maximum of 4 subjects will be dosed in account for

withdrawal and dropouts.

Hence, a maximum of 38 subjects will be randomized and dosed. No subjects should be

replaced after administered with the study treatment.

If possible, a maximum of two additional standby subjects (Stand by-I, Stand by-II) will be

enrolled to replace any subject, who is withdrawn or dropped due to any reason prior to

administration of study medication in period-1.

7.4 Justification of the Sample Size

Based on the in-house study data [3], a maximum intra subject variability of coefficient of

variation (ISCV %) of 23.1 was observed for C<sub>max</sub> of Paroxetine. According to NOM-177-

SSA1-2013, section 8.5.1.1, the statistical power must not be less than 80%. Based on the

observed maximum ISCV% of 23.1% and assuming the test/reference ratio of 95%, the

inclusion of 34 subjects in the study is required to meet at least a statistical power of 80% at

5% level of significance to achieve the results within 80.00-125.00% for 2-way crossover

study.

Using the intra-subject variability and the expected test/reference ratio from above paragraph,

the sample size is estimated from the following equation:

 $n_i \ge 2 [t_{1-\alpha, n-2} + t_{1-\beta, n-2}]^2 [CV/(-ln(\theta_L) - (-ln(\theta)))]^2$  where  $\theta \le 1$ 

Sponsor Code: 212969




### Bioequivalence Pivotal Study Protocol of Paroxetine tablets 20 mg under fasting conditions.

α: Probability of Type I error (0.05)

 $\beta$ : Probability of Type II error (0.1)

CV: Intra Subject Variability (0.231)

 $\theta$ : Expected T/R ratio (0.95)

 $\theta$ L: Lower bioequivalence limit (0.80)

Assuming the minimum sample size required (n) as 12, the sample size is estimated as follows:

$$n_i \ge 2 \left[ t_{1-0.05, \ 12-2} + t_{1-0.1, \ 12-2} \right]^2 \left[ 0.231 / \left( -\ln \left( 0.8 \right) - \left( -\ln \left( 0.95 \right) \right) \right]^2 \right]$$
 $n_i \ge 37$ 

Using the estimated sample size form previous iteration (n=37) from the above estimation, the sample size is again estimated as follows:

$$n_i \ge 2 \left[ t_{1-0.05, 37-2} + t_{1-0.1, 37-2} \right]^2 \left[ 0.231 / \left( -\ln \left( 0.8 \right) - \left( -\ln \left( 0.95 \right) \right) \right]^2$$
 $n_i \ge 32$ 

Using the estimated sample size form previous iteration (n=32) from the above estimation, the sample size is again estimated as follows:

$$n_i \ge 2 \left[ t_{1-0.05, 32-2} + t_{1-0.1, 32-2} \right]^2 \left[ 0.231 / \left( -\ln \left( 0.8 \right) - \left( -\ln \left( 0.95 \right) \right) \right]^2$$
 $n_i \ge 33$ 

Using the estimated sample size form previous iteration (n=33) from the above estimation, the sample size is again estimated as follows:

$$n_i \ge 2 \left[ t_{1\text{-}0.05, 33\text{-}2} + t_{1\text{-}0.1, 33\text{-}2} \right]^2 \left[ 0.231 / \left( -\ln \left( 0.8 \right) - \left( -\ln \left( 0.95 \right) \right) \right]^2$$

$$n_i \ge 33$$

Convergence has reached and the estimated sample size is at least 34 (round to equal number) subjects to meet at least a statistical power of 80% at 5% level of significance to achieve the results within 80.00-125.00% for 2-way crossover study.

### 7.5 Washout Period

There will be a washout period of at least 7 days between successive dosing.


> CONFIDENTIAL Avant Santé Research Center S.A. de C.V



Bioequivalence Pivotal Study Protocol of Paroxetine tablets 20 mg under fasting conditions.

## 7.6 Duration of the Study

The expected duration of the subjects' participation in the study will be at-least 12 days, including a wash-out period of 7 days between each dosing.

#### 7.7 Randomization

The order of receiving the test and reference products for each subject during each period of the study will be determined according to a randomization, generated by using SAS® software (version 9.4 or higher). This randomization will be balanced for the test product (A) and reference product (B). All the subjects should be divided into blocks of equal size and two-sequence "AB" and "BA" will be used for assignment of treatment in the respective study period (refer Figure-2). Analysts will not have access to the period randomization schedule. Randomization will be performed according to the procedure PB009 (Procedure for Randomization Schedule Generation).

# 7.8 Blinding

This study is an open label study; the subjects and the investigators will not be blinded towards the identity of the study treatments. Analysts (bioanalytical personnel) will be blinded with regard to the sequence of administration of test and reference products.

### 7.9 Test and Reference Products

**Table 3 Investigational Product Details** 

| IP Details | Reference Product (B) | Test Product (A) |
|---------------------|--------------------------|--------------------------|
| Distinctive Name | PAXIL | N/A |
| Generic name | Paroxetine hydrochloride | Paroxetine hydrochloride |
| Pharmaceutical form | Tablets | Tablets |
| Formulation | Immediate release | Immediate release |
| Strength | 20 mg | 20 mg |


Sponsor Code: 212969




Bioequivalence Pivotal Study Protocol of Paroxetine tablets 20 mg under fasting conditions.

| IP Details | Reference Product (B) | Test Product (A) |
|---|---|---|
| Dose | 20 mg | 20 mg |
| Lot / Batch No. (1) | To be designated | To be designated |
| Expiry date / Retest date (1) | To be designated | To be designated |
| Storage<br>Conditions | Store at 25°C (77°F): excursions permitted to 15–30°C (59–86°F). | Store at 25°C (77°F): excursions permitted to 15–30°C (59–86°F). |
| | | Manufactured by: |
| | | GlaxoSmithKline |
| Name of the | GlaxoSmithKline México, S.A. | Pharmaceuticals S.A. |
| manufacturer | de C.V. | Manufactured for: |
| | | GlaxoSmithKline México, S.A. |
| | | de C.V. |
| Sanitary<br>Registration<br>Number | 008M93SSA | Not applicable (2) |

<sup>1:</sup> Research Ethics Committee and Research Committee shall be notified on the lot / batch number and the expiry/retest date of the study drugs before conducting the clinical stage. The same information shall be notified to COFEPRIS in the final report of the study.

### 7.10 Reception and Storage of Investigational Products

In accordance to the NOM-177-SSA1-2013, a sufficient quantity of the investigational products (test and reference) will be supplied to the research center by the sponsor in its original marketing package (applicable for reference product) or in a sealed package along with its Certificate of Analysis (CoA) for the conduct of the study as well as for retention (once the study is completed). Therefore, at least 80 tablets of reference product and 80 tablets of test product will be supplied and stored at Avant Santé facilities, in order to guarantee the


<sup>2:</sup> The Test drug will be evaluated for obtaining COFEPRIS registration.



Bioequivalence Pivotal Study Protocol of Paroxetine tablets 20 mg under fasting conditions.

necessary resources for dosing the product of investigation at least once and also for its

retention (once the study is concluded to be able to repeat the study).

The study drug reception, handling and storage of investigational products will be performed

according to SOP CP017 (Study Drug Reception and Storage).

The test and reference products will be supplied in sealed packages.

Once received, both investigational products (test and reference) will be kept in separate

boxes (labeled with project number, IP name, IP type, batch number, manufacturing date and

/ or expiration date, and storage conditions along with "For clinical research use only"

statement) and stored in pharmacy as per the storage conditions mentioned on the label.

If the aforementioned conditions are not specified, the IPs will be stored as per the conditions

specified by the sponsor or the available literature.

Upon completion or termination of the study, the investigational products will be stored in

Avant Santé Research Center, S.A. de C.V. for at least 1 year after completion of the study or

until test product / reference product expiry date is due, whichever occurs first. Test and

reference products return or disposal will be followed according to respective in-house

procedures. [6,7]

• The test and reference products shall be in the valid expiry date at the time of the study

conduction.

• The percentage of assay content of the test product must be within the limits established

in the relevant pharmacopeias and it should not differ by more than 5% with that of the

reference product.

Criteria for acceptance or rejection of drugs are followed according to SOP CP017 (Study

Drug Reception and Storage).


Sponsor Code: 212969




Bioequivalence Pivotal Study Protocol of Paroxetine tablets 20 mg under fasting conditions.

7.11 Accounting of Investigational Products

The recording of the total quantity of investigational products received, dispensed, used,

retained, disposed or returned to the sponsor, will be performed in the respective forms and

kept in the pharmacy of Avant Santé Research Center, S.A. de C.V. The investigational

products balance will be included in the clinical study report. This activity will be performed

according to SOPs CP018 (Study Drug Dispensing and Retention) and CP019

(Investigational Products Return or Disposal).

7.12 Dispensing

The pharmacist will dispense required units of the test and reference products at least a day

prior the dosing in each period of the study under the supervision of a person from Clinical

Pharmacology department and a person from Quality Assurance. The doses will be transferred

to the dispensing containers as per the randomization schedule and properly labeled with the

project number, period number, subject number, IP type (test/reference) and storage

conditions, along with the following statement: "For clinical research use only".

At least one dose of each test and reference product will be dispensed as "standby" in order

to handle any unexpected loss or damage of the medications during their administration. This

activity will be performed according to CP018 (Study Drug Dispensing and Retention)

The test and reference product tablet will be removed from blister pack / package only at the

time of dosing.

Sponsor Code: 212969




Sponsor Code: 212969

Format No.: CPF127-03E No. Reference SOP: CP006

Bioequivalence Pivotal Study Protocol of Paroxetine tablets 20 mg under fasting conditions.

### 8.0 SELECTION AND WITHDRAWL OF SUBJECTS

# 8.1 Screening (selection and enrollment)

Healthy adult male & female volunteers, light or non or ex-smokers, aged between 18 and 55 years (both inclusive), with a weight  $\geq 50.00$  kg, with a BMI between  $\geq 18.0$  and  $\leq 27.0$  kg/m<sup>2</sup> will be selected according to the inclusion and exclusion criteria.

All the subjects will have a medical history during the selection and enrollment process.

Volunteers shall be found healthy according to the physical examination (including vital signs assessment), normal laboratory test results and 12-lead ECG.

The physical examination findings, ECG and laboratory tests will be considered valid for a maximum period of 90 days prior to the dosing on the first period of the study.

Pregnancy test in urine will be carried out during the screening period and at the time of each period check-in for all female subjects.

The process of selection and enrollment or withdrawal of subjects who will participate will be done according to the present protocol and as per the procedures CP002 (Volunteer Registration and Screening) and CP003 (Screening-Failing volunteers).

Real-time (RT-PCR) test for the detection and diagnosis of SARS-COV-2 will be carried out within the 72 hours prior to the first period check-in for all the subjects.

Avant Santé Research Center S.A. de C.V. will ensure the volunteer participation history by verifying the COFEPRIS database for bioequivalence studies.




Bioequivalence Pivotal Study Protocol of Paroxetine tablets 20 mg under fasting conditions.

#### **Clinical Laboratory Tests** 8.2

As part of the selection process the following laboratory tests will be performed to each subject.

**Table 4 Laboratory Tests** 

| Bloo | Urine analysis | |
|---|---|---|
| Hematology | Biochemistry | Office unarysis |
| Red blood cell count White blood cell count Differential white blood cell count Hemoglobin estimation Hematocrit Platelet count MCH, MCV, Mean Platelet Volume | Blood glucose (Random) Blood urea, Blood urea nitrogen (BUN) Serum creatinine Serum sodium, potassium and Chloride Serum uric acid Liver Function Tests: Total bilirubin Direct bilirubin Indirect bilirubin Blood glucose (Random) Protein Glucose Ketones Bilirubin Urobilinogen Blood / Red blood cells Nitrites Microscopic examination Pregnancy test (fer | |
| Serology HIV (1 & 2) antibodies HBsAg (Hepatitis B surface antigen) | SGOT (AST) SGPT (ALT) Serum alkaline phosphatase Total protein Serum albumin | Subjects) Urine drug screen Cannabinoids (Marijuana / Tetrahydrocannabinol- |
| HCV (Hepatitis C virus) antibodies) and VDRL | Serum Globulin<br>Lipid profile | THC), Cocaine, Opiates,<br>Amphetamine,<br>Methamphetamine and<br>Benzodiazepines |

Alcohol breath analysis test for all the subjects will be performed before check-in of each study period. Urine drug screen for all the subjects and pregnancy test in urine for female subjects will be performed before check-in of each period.

Real-time (RT-PCR) test for the detection and diagnosis of SARS-COV-2 will be carried out within the 72 hours prior to the first period check-in for all the subjects.

Project No./Protocol No.: AS/BK/OCT-19/0055  Version No: 02 (12/Oct/2020) Sponsor Code: 212969




Bioequivalence Pivotal Study Protocol of Paroxetine tablets 20 mg under fasting conditions.

# 8.3 Inclusion Criteria

Subjects must fulfill all of the following criteria to be considered for their inclusion in this study:

- 1. Healthy adult male or female subjects aged between 18 and 55 years (both inclusive).
- 2. Subjects is a light or non- or ex-smoker (A light\* smoker is defined as someone who smoke 9 or less cigarettes per day and an ex-smoker being defined as someone who completely stopped smoking for at least 6 months before day 1 of this study).
  - \*: If any subjects stop smoking during last 6 months before day 1 of the study and smoke 9 or less cigarettes per day, the subject will also be considered as a light-smoker.
- 3. With a weight  $\geq$  50.00 kg.

Sponsor Code: 212969

- 4. With a body mass index (BMI)  $\geq 18.0 \text{ kg/m}^2$  and  $\leq 27.0 \text{ kg/m}^2$ .
- 5. Found healthy according to the clinical laboratory results and physical examination (performed within 90 days prior to the dosing on period-1).
- 6. Have a normal 12 lead ECG and vital signs.
- 7. Have laboratory test results within the laboratory's stated normal range; if not within this range, they must lack of no clinical significance as judged by the PI or responsible physician.
- 8. Willing to avoid sexual contact or use an acceptable contraceptive method during the study including the washout period (for females). In case of male subjects, they should avoid sexual contact or use a latex or synthetic condom each time they have sex with a woman while taking Paroxetine and during 7 days after the end of the study.
- 9. If study subject is a female and is of child bearing potential, she shall practice a method of birth control for the duration of the study as judged by the investigator (s), like combined short acting (estrogen and progestogen containing) hormonal contraception e.g. oral, intravaginal, and progestogen-only hormonal contraception e.g. oral, intrauterine device




Bioequivalence Pivotal Study Protocol of Paroxetine tablets 20 mg under fasting conditions.

(IUD), intrauterine hormone-releasing system (IUS), condoms, foams, jellies and

diaphragm

Or

Abstinence

Or

If study subject is a female and is postmenopausal for at-least 1 year

Or

Is surgically sterile (bilateral tubal ligation, bilateral oophorectomy or hysterectomy has

been performed on the study subject).

10. Have a negative test for active COVID-19, within 72 hours prior to the first period check-

in. The testing should be done using a molecular (RT-PCR) approved by the country

regulatory authorities.

11. Subject is able to communicate effectively and voluntarily agreed to participate in this

study by signing written informed consent after being informed sufficiently about study

aspects like objectives, study procedures, characteristics of the investigational drug,

expected adverse events.

12. Subject willing to adhere to protocol requirements as described in informed consent

(written) approved by REC / RC.

8.4 Exclusion Criteria

Subjects will be excluded if they meet any of the following criteria:

a. If subject's age is less than 18 or older than 55 years.

b. Have any history of allergy or hypersensitivity to Paroxetine or to any of its

metabolites/derivatives or related drugs or excipients.

c. Have a positive test result for hepatitis B surface antigen (HBs Ag) or hepatitis C virus

antibody (HCV Ab) or HIV antibodies (types 1 and 2) or VDRL.


Sponsor Code: 212969




Bioequivalence Pivotal Study Protocol of Paroxetine tablets 20 mg under fasting conditions.

d. Subjects with symptoms suggestive of active COVID-19 infection (i.e. fever, cough,

respiratory difficulties) within 14 days of inpatient admission.

e. Subjects with known COVID-19 positive contacts\* within the past 14 days prior to the first

period check-in.

\*Positive Contact; this means, if the subject has been living, providing, care, being within

1.5 m for at least 15 min or having exposure to respiratory secretions with/to a person who

has COVID-19.

f. Study drug is contraindicated for medical reasons to the subject as per protocol section 3.7.

g. Have any history or presence of significant cardiovascular, pulmonary, hepatic, renal,

gastrointestinal, seizures, endocrine, dermatological, neurological or psychiatric disease or

disorder (e.g. Subjects with uncontrolled hypertension, phaeochromocytoma, carcinoid,

thyrotoxicosis, bipolar depression, schizoaffective disorder and acute confusional states).

h. Presence of significant gastrointestinal, hepatic or kidney disease, or surgery or any other

conditions known to interfere with the absorption, distribution, metabolism or excretion of

drugs or known to potentiate or predispose to undesired effects.

Or

Subjects with a history of gastrointestinal disorder or surgery which may affect the

absorption of investigational drug.

i. Have a history of alcohol abuse or drug abuse during the last 1 year prior to period-1

dosing.

j. Have a history of smoking  $\geq 10$  cigarettes per day during the last 6 months prior to period-

1 dosing.

k. Have history or presence of cancer.

1. Have any history of gastrointestinal ulcers / intestinal bleeding.

m. Have difficulty in swallowing solid medications such as tablet.

n. Have history of difficulty for donating blood.


Sponsor Code: 212969




### Bioequivalence Pivotal Study Protocol of Paroxetine tablets 20 mg under fasting conditions.

- o. Have clinically significant abnormal laboratory tests results.
- p. Have a systolic blood pressure < 90 or > 140 mmHg or diastolic blood pressure is < 60 or > 90 mmHg.
- q. Have a pulse rate < 60 beats/minute or > 100 beats/minute (Lower range of pulse range will be accepted up to 45 beats/minute in case of athlete).
- r. Have used any prescribed medication during the last 14 days preceding the first dosing, or use OTC, medicinal or herbal products during the last 7 days or use medicinal enzyme inhibitors / inducers during last 30 days preceding the first dosing.
- s. Have participated in a drug research study or donated blood within the last 3 months.
- t. Have a positive result for drugs of abuse test [Cannabinoids (Marijuana/Tetrahydrocannabinol-THC), Cocaine, Opiates/Morphine, Amphetamine, Methamphetamine and Benzodiazepines] performed during screening.
- u. Female subject, who is currently breast feeding or a who is pregnant or who is likely to become pregnant during the study.
- v. Female subject has a positive pregnancy test results.
- w. Unwillingness or inability to comply with the instructions on the lifestyle described in this Protocol.
- x. If the PI considers, for any reason, that the volunteer is not a suitable candidate to receive the study drug.

### 8.5 Criteria for Subject Withdrawal from the Study

Sponsor Code: 212969

Subjects have the right to withdraw their consent from the study at any time and for any reason without facing any related prejudice. The Principal Investigator may withdraw a subject from the study if:




Bioequivalence Pivotal Study Protocol of Paroxetine tablets 20 mg under fasting conditions.

a. The subject wishes to withdraw consent (In case the subject request to disposal of the

collected samples, the same shall be documented and will be informed to sponsor and

REC/RC).

b. The subject suffers from significant inter-current illness or undergoes surgery during the

study. In case a subject is positive for COVID-19 or has a related symptom (i.e. fever,

cough, respiratory difficulties), they shall be isolated for 14 days and they shall be

discontinued In case any other subject was exposed to a COVID-19 patient, they must

report this to Avant Santé, GSK and/or their primary care provider.

c. Subject fails to comply with the requirements of the protocol section 9.3 Restrictions.

d. Subject experiences an adverse event and it is not in the subject's best interest to continue

in the study (as judged by the PI).

e. Subject has a positive result for the breath alcohol test or urine drugs of abuse test

[Cannabinoids (Marijuana/Tetrahydrocannabinol-THC), Cocaine, Opiates/Morphine,

Amphetamine, Methamphetamine and Benzodiazepines] prior to check-in of each study

period.

f. The subject vomits at the time of the drug administration or vomiting / diarrhea occurs

within 10 hours of drug administration (representing twice the median  $T_{max}$  of 5 hours).

g. In case of a female subject a positive result for the pregnancy test.

h. Subjects who miss 4 or more consecutive blood draws in any of the study periods.

According to NOM-177-SSA1-2013, section 8.9.5, frequent sampling points are needed

around the T<sub>max</sub> and also at least four samples during the log-terminal phase to obtain the

extraction rate constant. If any subject misses 4 or more consecutive sampling points during

the absorption phase or the extraction phase, it will have an impact on the precise accuracy

of the C<sub>max</sub> and AUC curve.

i. The study is suspended or terminated by the sponsor or PI or EC/REC.




Bioequivalence Pivotal Study Protocol of Paroxetine tablets 20 mg under fasting conditions.

It should be noted that any subject that is not discontinued or withdrawn from the study will be considered as a subject who finishes the study.

9.0 TREATMENT OF SUBJECTS

9.1 Drug Administration

In each study period, all subjects will be required to fast overnight for at least 10.00 hours prior to dosing until at least 04.00 hours post-dose.

In each study period, a single-dose of either the test product (A) or reference product (B) will be orally administered to the subjects in sitting posture along with 250 mL of water at room temperature under fasting conditions.

The administration of the test or reference products to each subject will be performed as per a randomization schedule.

The subjects will be instructed to swallow the tablet as a whole as mentioned in the prescribing information and not to touch the tablet with their hands, chew or crush the tablet since this can affect the drug release.

Subject's hands and mouth will be checked after dosing to ensure compliance with dosing.

Immediately after dosing in each period trained study personnel will evaluate the compliance by supervising the complete administration procedure (SOP CP020, Administration of the Investigational Product).

Drug administration will be registered in the respective source documents.

9.2 Dietary Plan

Subjects will be provided with standard meals throughout their stay in the facilities.

On the check-in day (day -1) they will receive dinner, which will be finished at the latest 10.00 hours prior to dosing at the following day in each study period.

Subjects will be required to fast overnight for at least 10.00 hours prior to dosing and until at least 04.00 hours post-dose in each study period.


Sponsor Code: 212969




### Bioequivalence Pivotal Study Protocol of Paroxetine tablets 20 mg under fasting conditions.

After the dose administration of test or reference product (day 1), lunch, snack and dinner will be provided at 04.00, 08.00 and 12.00 (with a grace period of + 45 minutes) hours post-dose respectively, in each study period.

The meal plan will be uniform for all the subjects and same between the study periods.

Information on the amount of meal consumed and the time of consumption by each subject will be registered in the respective source documents. The nutritional value of the meals is presented in the following table.

Table 5 Nutritional value of diet on study day 1

| Nutritional Value of meals | |
|----------------------------|--------------|
| 2000 kcal ± 10% | Calories (%) |
| Proteins | 15-20% |
| Lipids | 25-30% |
| Carbohydrates | 50-60% |
| Total | *100% |

<sup>\*%</sup> of kilocalories is within its adequate distribution of 90–110%.

#### 9.3 Restrictions

# **Smoking**

All subjects will be instructed to refrain from smoking of cigarettes / nicotine containing products for at least 72.00 hours prior to the dosing and until the last sample collection in each period and will be prohibited from smoking during their in-house stay.

### **Medications**

Sponsor Code: 212969

All subjects will be asked about their medication history. They will be instructed not to take any medication until the study is completed; particularly during the last 14 days preceding the first dosing for any prescribed medication, the last 7 days before for OTC medicinal or herbal products used for therapeutic purposes, and the last 30 days before for any enzyme inhibiting / inducing drugs preceding the first dosing.




Bioequivalence Pivotal Study Protocol of Paroxetine tablets 20 mg under fasting conditions.

Subjects will be specifically reminded that the restriction mentioned above includes

analgesics, cold & anti-allergic preparations, vitamins and natural products used for

therapeutic benefits and antacid preparations.

Vitamins used as nutritional supplements in non-therapeutic doses (as judged by the principal

investigator or designee) may be accepted, but their consumption must be stopped from at

least 7 days prior to the dosing and until the study is completed.

If a drug therapy other than that specified in the protocol is required prior to, during the study

or in the washout period, the Principal Investigator shall decide whether to continue or

discontinue the subject's participation based on the following:

The pharmacology and pharmacokinetics of the non-study medication.

> The likelihood of a drug-drug interaction, which may affect the pharmacokinetic

comparison of the study drugs.

The time and duration of administration of the non-study medication.

• Diet

All subjects will be instructed to avoid the consumption of any xanthine-containing food or

beverages (tea, coffee, theobromine, theophylline, chocolates, cola drinks, etc.) at least 72.00

hours prior to the dosing and until the last blood sample collection in each study period.

Subjects will be instructed to avoid the consumption of alcohol (or related products) as well

as smoked or carbon cooked food from at least 72.00 hours prior to the dosing, until the last

blood sample collection in each study period.

Subjects will be instructed to avoid the consumption of pomelos or grapefruit juice or products

containing grapefruit extract (e.g. soda) from at least 72.00 hours prior to the dosing, and till

the last blood sample collection in each study period.

The consumption of above-mentioned products will also be prohibited during their in-house

stay.

Sponsor Code: 212969




Bioequivalence Pivotal Study Protocol of Paroxetine tablets 20 mg under fasting conditions.

Fluid (water) restriction

The subjects will not be allowed to drink water 1 hour before and until 2 hours post-dose except for the 250 mL of water provided for the dosing, unless it is clinically indicated; at all

other times water will be provided ad libitum.

Postural (activity) Restriction

The dose will be administered to all subjects at the scheduled time and subjects will be instructed to remain in comfortable sitting position for the first 02.00 hours following the drug

administration except when clinically indicated or protocol specified activity (blood sample

collection) or due to natural exigencies.

After 02.00 hours post-dose, subjects will be allowed to wander and will be advised to avoid

any severe physical exertion.

In case of an adverse event (AE), subjects will be maintained in the proper position as per

physician's assessment in each study period.

Recommendations during washout period and visits to the center (ambulatory samples)

In case a subject has symptoms of COVID-19, the following recommendations will be

provided (the same as dictated by the WHO):

• Isolation for 14 days at home: Staying at home except to get medical care immediately

if having an emergency warning sign (i.e., trouble breathing).

• Monitoring temperature: average human body temperature is 36-37°C.

Any related-COVID-19 symptom, worsening or recovery, must be reported to their

primary care provider and to Avant Santé Principal Investigator.

9.4 Housing

Sponsor Code: 212969

Subjects will be in the clinical facility from at least 10.50 hours prior to the dosing until the

last in-house blood sample collection i.e. 24 hours in each study period.

Subjects will visit clinical facility at 36.00, 48.00 and 72.00 hours for the collection of the

ambulatory samples in each study period.




#### Bioequivalence Pivotal Study Protocol of Paroxetine tablets 20 mg under fasting conditions.

Subjects will be instructed to self-quarantine during the outpatient period of the study i.e. until 72 h blood sample collection in period-2 or until withdrawal, whichever is earlier, and to monitor at home their daily body temperature.

# 9.5 Sampling Schedule

In each study period, a total of 24 blood samples (4 mL each) will be collected from each subject as per the following schedule:

- The first blood sample will be collected within 1.50 hours prior to the dosing (00.00 hours / pre-dose).
- The remaining samples will be collected after the dosing of the test or reference drug at 00.50, 01.00, 01.50, 02.00, 02.50, 03.00, 03.50, 04.00, 04.50, 05.00, 05.50, 06.00, 06.50, 07.00, 08.00, 09.00, 10.00, 12.00, 16.00, 24.00, 36.00, 48.00 and 72.00 hours.
- The samples corresponding to 36.00, 48.00 and 72.00 hours post dose will be collected on separate visits as ambulatory sample in each period of the study.

The total blood volume collected from each subject will not exceed 223 mL, which includes about 10 mL for the selection process (selection and enrollment), 21 mL for the discarded heparinized blood and 192 mL for the pharmacokinetic evaluation.

If circumstances arise, where more than 223 + 10 mL (may be collected for safety evaluation purpose) of blood from each subject needs to be withdrawn the subject will be asked for additional consent and the REC / RC will be informed.

Table 6 Blood volume of samples to be collected during the study

| Sample Type | Sample | Number of Sampling Times | | | Total Volume |
|---|---|---|---|---|---|
| затри турс | Volume (mL) | Screening | Study Period | Follow-Up | (mL) |
| Screening | 10 mL | 1 | | | 10 |
| PK Blood<br>Samples | 4 mL | | 48 samples<br>(Period 1,2) | | 192 |
| Heparinized blood | 0.5 mL | | 42 samples<br>(Period 1,2) | | 21 |


Sponsor Code: 212969




Bioequivalence Pivotal Study Protocol of Paroxetine tablets 20 mg under fasting conditions.

**TOTAL** 223

At the time of each blood sample collection, 4 mL will be collected through an indwelling cannula placed temporarily (for at least 24.00 hours post-dose) in a forearm vein or as per subject's convenience for practical reasons and the remaining sample(s) will be collected through direct venipuncture.

Blood samples will be obtained in K<sub>2</sub>-EDTA vacuum tubes (pre-labeled with project number, period number, subject number and sample number).

If the times of sample collection vital signs or medical examination and food consumption overlap during the housing period, the order will be as follows.

Sample collection  $\rightarrow$  vital signs or medical examination  $\rightarrow$  food consumption.

Blood samples shall be collected not earlier or later than (±) 2 minutes of the specified sampling time for all the in-house samples and not earlier or later than  $(\pm)$  60 minutes of the specified sampling time for ambulatory samples. Blood sampling will be registered in the respective source documents.

If blood samples are collected earlier or later than this period from the scheduled time, this shall be reported as a deviation from this protocol.

Heparin-lock technique (with 0.5 mL) will be used to prevent coagulation of the blood in the cannula. Prior to the blood collection through the cannula, 0.5 mL of heparinized blood will be withdrawn and discarded in order to prevent the heparin interfering with the sample analysis. If for any reason the indwelling cannula is blocked or removed, direct venipuncture will be performed to collect the samples.

All this process is described in detail in the procedure CP021 (Phlebotomy Performance).

If any subject misses any blood sampling point, it will be considered as missing sample.

The same will be denoted as (M), it will be considered as protocol deviation and mentioned in the clinical study report.




Bioequivalence Pivotal Study Protocol of Paroxetine tablets 20 mg under fasting conditions.

9.6 Sample Processing and Storage

Once collected, the blood samples will be placed in an ice-filled container or another cooling

device until the centrifugation process is started.

Centrifugation process will be started within 45 minutes from the time of blood sample

collection and will be performed at 3000 rpm for 10 minutes at  $4 \pm 2$  °C.

The plasma obtained from blood samples will be transferred as soon as possible into two

different cryo-tubes (aliquot 1 and aliquot 2), pre-labeled with project number, period number,

subject number, sample number and aliquot number.

The plasma volume obtained from blood sample will be allocated as follows:

Aliquot 1: 1.0 mL of plasma (approximately).

Aliquot 2: rest of the plasma.

All plasma samples (aliquot 1 for sample analysis and aliquot 2 as back-up) will be stored in

the Clinical facility at a temperature of -50 °C or below until transferred in dry ice to the

Bioanalytical facility, where they will be stored at a temperature of -50 C or below until their

analysis.

9.7 Sample transfer

At the end of each period or clinical phase, samples will be separated and sorted by subject,

period and aliquot as per the procedure CP031 (Biological Samples Processing, Storage,

Shipment and Spillage Handling). Once the samples of each subject are sorted, they will be

placed in propylene storage containers or in an auto-sealed bag, previously labeled with the

project number, period number, subject number, aliquot number and number of samples.

Process of separation, sorting and sample verification will be done with sufficient dry ice.

Temperature will be monitored during the separation sorting and verification process with a

calibrated data-logger and under supervision of quality assurance department personnel.

At the end of the clinical phase of the study or each study period, aliquot 1 (used for the

quantification and re-analysis) samples will be shipped for analysis to the Bioanalytical




Bioequivalence Pivotal Study Protocol of Paroxetine tablets 20 mg under fasting conditions.

facility in a container with dry ice while transfer and temperature will be monitored. The

aliquot 2 (for back-up) samples will be shipped using the same procedure and only after

confirming the reception or loss of the aliquot 1 samples. If required, Aliquot 2 will be used.

Aliquots will be stored in different deep freezers under the same condition in bioanalytical

area.

The process of reception, handling, storage and disposal of biological samples in the

Bioanalytical unit, will be carried out according to procedure BL021 (Reception,

Management, Storage, Transfer and Disposition of Biological Samples).

CP personnel shall send the information "subjects samples to be analyzed" (including the

reason or justification for not analyzing other samples of subjects) to the Bioanalytical

department with the approval of the Principal Investigator and authorized by QA.

10.0 ASSESSMENT OF EFFICACY

As this is a bioequivalence study, no efficacy assessment will be performed. The

pharmacokinetic parameters of the test and reference formulations will be assessed.

11.0 ASSESSMENT OF SAFETY (CLINICAL SAFETY MEASURES)

11.1 Recording of Vital Signs and Medical Examination

Medical examination, which consists on subject's anamnesis, inquiry for possible AEs,

evaluation of vital sings and overall health status to determine if further physical examination

is required will be performed before check-in, prior to the dosing and before the check-out in

each study period.

Nevertheless, it may also be performed at any time during the study conduction if judged

necessary by the physician.

Physical examination, which consists on subject's anamnesis, examination of the head, neck,

thorax, abdomen, and extremities (but not limited), inquiry for possible AEs and evaluation




Bioequivalence Pivotal Study Protocol of Paroxetine tablets 20 mg under fasting conditions.

of vital sings will be performed before check-in of each study period and may also be

performed at any time during the study conduction if judged necessary by the physician.

Vital signs (sitting blood pressure, pulse rate, respiratory rate and axillary body temperature)

will be measured and registered before check-in, prior to dosing, at 03.00, 05.00 and 12.00

hours (within ±45 minutes) hours after the dosing, before the check-out and at the time of

each ambulatory sample collection in each study period.

The subjects' well-being (assessed by verbal questionnaire to gather information about AEs)

will be asked at the time of the medical examination, during the vital signs recording and at

the time of each ambulatory sample collection in each study period; this will be registered in

the respective source document.

Seven (7) to 9 days after the collection of 72-h blood sample in second period or after the

withdrawal, a telephone call will be made to each subject by the personnel designated by the

PI to monitor any serious adverse event, specifically, subjects will be questioned about any

symptoms related to COVID-19.

11.2 Identification, Handling and Reporting of AE and SAE

Definitions

Adverse Event (AE): Any untoward medical occurrence that may occur in a research subject

during the clinical research phase of a drug or vaccines but which does not necessarily has a

causal relationship with this.

An adverse event can therefore be any unfavorable and unintended sign (including an

abnormal laboratory finding), symptom, or disease temporally associated with the use of a

drug (research product), whether or not considered related to the research product.

Abnormal laboratory results will be reported as adverse events under the following

circumstances:

• When the abnormal lab report is accompanied with associated symptoms.




Bioequivalence Pivotal Study Protocol of Paroxetine tablets 20 mg under fasting conditions.

• When a medical or surgical intervention is required.

• When an additional diagnostic test is required.

• When it precedes and is associated with any of the outcomes included in the definition of

serious adverse event.

• When it is so considered by the PI.

• Abnormal laboratory value as well as a significant shift from baseline within normal range

which the qualified investigator or medically qualified delegate considers to be clinically

significant (CS). If the Principal Investigator or the qualified medical delegate considers

the abnormalities to be not Clinically Significant (NCS), the abnormalities do not need to

be reported as AE.

Therefore, a clinically significant laboratory value is one that indicates a new disease process,

exacerbation or worsening of an existing condition or that requires additional measures.

Adverse Drug Reaction (ADR): Any undesirable effect, associated with the use of a drug that

may occur as part of the drug's pharmacological action or may be unpredictable in its

occurrence.

Suspected Adverse Drug Reaction (SADR): Any unwanted clinical manifestation that gives

an indication or appearance of having a causal relationship with one or more drugs.

Unexpected Adverse Drug Reaction (UADR): an adverse reaction which nature or severity

is not described in scientific literature, neither in the label nor in the applicable product

information, nor in the documentation presented for its registration, additionally, that it is not

possible to infer it from its pharmacological activity and that it may be more serious that

indicated on the label.

<u>Serious Adverse Event (SAE)</u>: any medical occurrence that at any dose:

• Put patient's life in risk or results in death.




Bioequivalence Pivotal Study Protocol of Paroxetine tablets 20 mg under fasting conditions.

• Requires in-patient hospitalization or prolongation of existing hospitalization.

• Results in persistent or significant disability/incapacity.

• Is a congenital anomaly/birth defect.

• Other important medical events: events that may not be immediately life-threatening or

result in death or hospitalization, but may jeopardize the patient or may require

intervention to prevent one of the other outcomes listed in the definition.

Identification of Adverse Events

The subjects will be monitored throughout the study for any adverse event manifestation.

They will be encouraged to report any sign, symptom, and any health change to the clinical

staff. The severity of each AE and its relationship to the study treatments will be determined

by the PI based on observation and questioning of the subjects and in accordance to the

following classification: non-assessable or unclassifiable, conditional or unclassifiable,

unlikely, possible, probable or certain.

The following measures will be employed to ensure that the adverse event is detected at the

earliest:

• The physical examination and vital signs recording will be performed at regular intervals

after the study drug administration.

• The subjects' well-being will be enquired at regular intervals (see section 11.1).

• All subjects who have received at least a single dose of the study drug will undergo a

complete medical evaluation after the completion of the last sample collection for safety

reasons.


Sponsor Code: 212969




Bioequivalence Pivotal Study Protocol of Paroxetine tablets 20 mg under fasting conditions.

• Management of Adverse Events

A medically qualified designee will be available round-the-clock during the period of housing

at the clinical facility. If any subject develops an AE the following measures will be adopted:

• Subject will be evaluated by the physician or designated personnel, treated and/or

followed-up until the symptoms disappear or laboratory values return to normal levels, as

judged by the PI.

• In case of a SAE, subject will be treated by a physician in the ICU, fully equipped with all

the emergency handling material like defibrillator, ventilation mask, ECG machine,

suction apparatus, etc., or may be referred to the contract hospital.

Recording of Adverse Events

Any symptom, sign or significant abnormal laboratory finding (after repeat test confirms the

abnormality) whether observed or reported during the course of the study (i.e., within 7 to 9

days after the last sample collection or after the withdrawal) will be recorded as an adverse

event whether it has a causal relationship with the drug or not.

The following information has to be individually recorded for each AE in an Adverse Event

reporting form:

• Description of the AE.

• Subject number, period, date and time of last dosing.

• Type of adverse event.

• Seriousness of adverse event.

• Date and time of onset/reporting.

• Date and time of resolution.

• Intensity (mild, moderate or severe).



No. Reference SOP: CP006 Format No.: CPF127-03E

### Bioequivalence Pivotal Study Protocol of Paroxetine tablets 20 mg under fasting conditions.

- Relatedness to the study medication (non-assessable or unclassifiable, conditional or unclassifiable, unlikely, possible, probable or certain).
- Action taken or treatment given.
- Outcome of adverse event (resolved or unresolved).
- Follow-up.
- Further details of the AE (if any).

Severity (Intensity) of the adverse event, adverse reaction suspicion and adverse reactions, will be classified according to the clinical manifestation as:

Mild: Signs and symptoms easily tolerable, which do not need treatment, do not prolong hospitalization and do not require medicine product suspension.

Moderate: Interferes with usual activities (may cause work or school casualties), without directly threatening the patient's life. It requires pharmacological treatment and may or may not require the suspension of the causative drug.

Severe: Interferes with usual activities (may cause work or school dropouts). It requires pharmacological treatment and the suspension of the causative drug.

Adverse reactions are classified according to the assessment of causality as (see table 7):

**Table 7 Adverse Reaction Classification** 

| Causality<br>Term | Assessment Criteria |
|---|---|
| Certain | <ul> <li>Clinical event, including alterations in laboratory tests, which manifests itself with a plausible temporal sequence in relation to the administration of the drug.</li> <li>It cannot be explained by the concurrent disease, or by other drugs or substances.</li> <li>The response to drug suppression (withdrawal) must be clinically plausible.</li> </ul> |




Sponsor Code: 212969

Format No.: CPF127-03E No. Reference SOP: CP006

Bioequivalence Pivotal Study Protocol of Paroxetine tablets 20 mg under fasting conditions.

| Causality<br>Term | Assessment Criteria |
|---|---|
| | • Event shall be definitive pharmacologically or phenomenological, using, if necessary, a conclusive re-exposure procedure. |
| Probable | <ul> <li>Clinical event, including alterations in laboratory tests, which manifests itself with a reasonable temporal sequence in relation to the administration of the drug.</li> <li>Unlikely to be attributed to the concurrent disease or by other drugs or substances, and that when the drug is withdrawn, a clinically reasonable response is presented.</li> <li>It is not required to have information on re-exposure to assign this definition.</li> </ul> |
| Possible | <ul> <li>Clinical event, including alterations in laboratory tests, which manifests itself with a reasonable temporal sequence in relation to the administration of the drug.</li> <li>Could also be explained by the concurrent disease or by other drugs or substances.</li> <li>Information on drug withdrawal may be lacking or unclear.</li> </ul> |
| Unlikely | <ul> <li>Clinical event, including alterations in laboratory tests, manifested with an unlikely temporal sequence in relation to the administration of the drug.</li> <li>It could be explained more plausibly by the concurrent disease, or by other drugs or substances.</li> </ul> |
| Conditional /<br>Unclassifiable | • Clinical event, including alterations in laboratory tests, reported as an adverse reaction, from which it is essential to obtain more data in order to make an appropriate evaluation, or additional data are under examination. |




No. Reference SOP: CP006 Format No.: CPF127-03E

Bioequivalence Pivotal Study Protocol of Paroxetine tablets 20 mg under fasting conditions.

| Causality<br>Term | Assessment Criteria |
|---|---|
| Unassessable /<br>Unclassifiable | Notification that suggests an adverse reaction, but that cannot be judged because the information is insufficient or contradictory and cannot be verified or completed with provided data. |

# Reporting of non-serious Adverse Events / non-serious Adverse Drug Reactions

All non-serious, ADRs (expected or unexpected) and AEs occurred during the study conduction shall be notified to the REC/RC and the sponsor by the PI in the final study report according to SOP CP025 (Adverse Events and Serious Adverse Events Recording, Monitoring and Reporting).

# Reporting of Serious Adverse Events / Serious Adverse Drug Reactions

All SAEs and SADRs shall be reported immediately (within the first 24 hours after their occurrence) to the REC/RC, Sanitary Responsible and Sponsor's responsible person either by telephone or written form.

The information to the sponsor shall be sent in attention to:

PPD

GlaxoSmithKline México, S.A. de C.V. Calzada México Xochimilco No. 4900

Col.San Lorenzo Huipulco 14370 Ciudad de México

Phone number: PPD

Email: PPD

Sponsor Code: 212969

The event must also be documented on the "Adverse Event" section in the CRF and in the clinical report. All SAEs must be transcribed in the CRF, whether or not there is a causal relationship with the drug or medicinal product being evaluated.




Bioequivalence Pivotal Study Protocol of Paroxetine tablets 20 mg under fasting conditions.

The regulatory authorities (CNFV) shall be notified according to what is established in the

"Pharmacovigilance guide for the notification of AE, SADR, ADR, and ESAVI or any safety

problem related to the use of drugs" and according to the NOM-220-SSA1-2016, through the

platform assigned by the CNFV for this purpose and in the Final Safety Report.

The notification through the platform assigned by the CNFV for this purpose shall be

performed according to the timelines stablished in the valid NOM-220-SSA1-2016.

Notification to the CNFV of serious adverse events will be made by Avant Santé, using the

current MedDRA terminology. [7-10]

Actions to be taken if Pregnancy Occurs

If a female subject becomes pregnant during their participation in the clinical study, she will

be immediately withdrawn from the study and will be monitored throughout the pregnancy

to assess drug AEs and ADRs in the mother / fetus or infant. The investigator must inform

the Sponsor's safety division within 24 hours after being aware of a confirmed report of

pregnancy fulfilling any of the following criteria:

> Reports of congenital anomaly(ies) in fetus, child,

> Reports of spontaneous abortion,

Reports of late fetal death,

Reports of ADRs in new born / neonate that is fatal, life threatening, resulting in persistent

or significant disability / incapacity or resulting in or prolonging hospitalization,

When the medicinal products are known (or suspected) to induce teratogenic or foeto-toxic

effects and are therefore contraindicated (or not recommended) in pregnant women, the

circumstances relating to the pregnancy must be documented (e.g. patient "not aware" of the

risk, contraception failure). Cases with all such drugs whether or not associated with any

congenital anomaly and / or serious adverse drug reaction must always be considered serious

and reported on expedited basis to regulatory authorities. Teratogenic potential of the drug

must be determined from the safety section of the literature.




#### Bioequivalence Pivotal Study Protocol of Paroxetine tablets 20 mg under fasting conditions.

All pregnancy reports not fulfilling the above criteria must be reported by the Principal Investigator at the earliest and no later than 3 working days of receipt of confirmed report of pregnancy.

The Principal Investigator/ Designated personnel will follow up and collect pregnancy information as per the following schedule to determine outcome including spontaneous or voluntary terminations, details of birth, presence or absence of congenital anomalies, and maternal or newborn complications etc.

Table 8 shows the follow-up schedule in case of pregnancies during the study.

Table 8 Pregnancy follow up

| No. | Follow up |
|-----|--------------------------------------------------------|
| 1 | Initial Contact |
| 2 | First Trimester (3 months Gestation) |
| 3 | Second Trimester (6 months Gestation) |
| 4 | Third Trimester (9 months Gestation) |
| 5 | At birth |
| 6 | 30 days after birth |
| 7 | 6 months after birth (In-case of congenital anomalies) |

The principal investigator / designee must obtain the minimum required information, with documentary evidence, if any, from the subject's Obstetrician / Gynecologist / Pediatrician.

# Follow-Up of Adverse Events

Sponsor Code: 212969

Classification of AE will be done by the PI, as well as causality relation. In case of SAE, causality will be confirmed by the sponsor (for test product).

Subjects will be instructed to report at the clinical facility for any AE during the washout period. All the adverse events will be treated by the PI or CI at the clinical facility or in the contract hospital. All AEs will be followed up wherever possible until their resolution or until the CI or PI believes that there will be no further changes. This may involve additional visits.




Bioequivalence Pivotal Study Protocol of Paroxetine tablets 20 mg under fasting conditions.

Follow-up and closure of adverse events will be done according to the procedure CP025

(Adverse Events and Serious Adverse Events Recording, Monitoring and Reporting).

12.0 **BIOANALYSIS** 

12.1 Sample analysis

The concentrations of Paroxetine in plasma samples will be quantified using a validated

bioanalytical UPLC/MS-MS method (LOQ - 0.106 ng/mL) according to COFEPRIS

guidelines, GLP and in-house SOPs.

Method validation and subject sample analysis will be performed using same the

anticoagulant (K<sub>2</sub>-EDTA) that will be used for blood sample collection in clinical phase.

The use of reference substances of Paroxetine and internal standard, calibration curve spiking

and control points as well as subject sample analysis shall be performed according to the

stability periods mentioned in the Method SOP and according to the procedure BL004

(Sample Analysis, Acceptance and Re-assay Analysis of Study Samples). Samples for

reanalysis and its acceptance shall be performed according to the procedure BL004 and the

cause of the same will be mentioned in the report.

Quality control samples will be distributed throughout each batch of the study samples

analyzed. The analyst will not have access to the randomization schedule, which is used for

dispensing.

12.2 Reporting of drug concentration data

After completion of the analysis, all the concentration data will be transferred to the

Pharmacokinetic and Biostatistics Department. All concentration values below the lower limit

of quantification (LLOQ) will be reported as BLOQ and any missing samples will be reported

as "NE".

If the pre-dose concentration is above LLOQ, then pre-dose concentration will be reported as

such for pharmacokinetic analysis.

Sponsor Code: 212969




Bioequivalence Pivotal Study Protocol of Paroxetine tablets 20 mg under fasting conditions.

All the concentration data should be reported in the bioanalytical report according to SOP:

BL018 (Preparation of sample analysis report).

Overall (mean) accuracy and precision of the QC samples of all accepted runs should be

calculated at each concentration level and reported in the bioanalytical report according to

SOP BL018 (Preparation of sample analysis report).

13.0 PHARMACOKINETIC PARAMETERS

Non-compartmental pharmacokinetic analysis will be performed on the observed plasma

concentration of Paroxetine using WinNonlin® software (6.4 version or higher).

Any concentration below lower limit of quantification (BLOQ) including pre-dose

concentrations will be converted to zero.

If the pre-dose concentration is  $\leq 5\%$  C<sub>max</sub> of the respective period and above LLOQ,

then pre-dose concentration will not be converted to zero and the respective subject shall

be considered for pharmacokinetic and statistical analysis.

Missing samples will be reported as "NE" and will not be included for pharmacokinetic and

statistical analysis. The process will be performed according to the procedure PB003

(Procedure for Statistical Analysis using WinNonlin).

The following pharmacokinetic parameters will be computed.

**Primary parameters** 

C<sub>max</sub> : Maximum observed concentration following each treatment.

The area under the concentration versus time curve from time  $AUC_{0-t}$ 

zero to the last measurable concentration using linear

trapezoidal linear interpolation method.


**Secondary parameters** 

 $T_{max}$ : Time of the maximum measured concentration.


Sponsor Code: 212969




#### Bioequivalence Pivotal Study Protocol of Paroxetine tablets 20 mg under fasting conditions.

The area under the concentration versus time curve from time

zero to infinity calculated; Where  $AUC_{0-inf} = AUC_{0-t} + C_t / \lambda z$ ,

AUC<sub>0-inf</sub> Ct is the last measurable concentration and  $\lambda z$  is the terminal

elimination rate constant.

The residual area in percentage  $[(AUC_{0-inf} - AUC_{0-inf})/AUC_{0-inf}]$ 

AUC % Extrap

x 100

First order rate constant associated with the terminal portion

of the curve (log-lineal). This is estimated via linear regression

Lambda z of time vs. log concentration. This parameter will be calculated

using at least three or more non-zero plasma concentration

values

The elimination half-life will be calculated as  $0.693/\lambda z$ HL Lambda  $z(t\frac{1}{2})$ 

#### Note:

Sponsor Code: 212969

For all the above computations, actual time points of the sample collection will be used in case of sample collection deviations i.e. beyond  $\pm 2$  minutes.

➤ No value of Lambda z (Kel), AUC<sub>0-inf</sub>, or HL Lambda z (t½) will be reported for cases who do not exhibit a terminal Log-linear phase in the concentration versus time profile.

> Statistical methods used in the study will be mentioned in the Statistical Analysis Plan.

#### 14.0 STATISTICAL ANALYSIS

 $(K_{el})$ 

Data from all treated subjects will be included in the statistical analysis.

If any of the subject's data is eliminated from the statistical analysis which meet the criteria of section 14.9 'Criteria for elimination of subject data from the statistical analysis', statistical analysis shall be performed and presented with and without the data of eliminated subject's data.




Bioequivalence Pivotal Study Protocol of Paroxetine tablets 20 mg under fasting conditions.

The statistical analysis will be carried out according to the PB005 procedure (Procedure for

Statistical Analysis for a cross-over design).

Statistical analysis of PK parameters for establishing bioequivalence will be performed using

the software SAS® (version 9.4 or higher). PROC GLM will be used for the estimation of the

geometric least square mean differences (test - reference) of the test and reference

formulations on the In-transformed PK parameters C<sub>max</sub> and AUC<sub>0-t</sub> for Paroxetine and the

corresponding standard errors of the differences will also be computed. Based on these

parameters, 90% confidence intervals will be constructed for the geometric least square mean

differences of In-transformed C<sub>max</sub> and AUC<sub>0-t</sub> for Paroxetine.

The anti-ln (or exponential) of the limits obtained from the ln-transformed data will give the

90% confidence interval for the ratio of geometric least square means of test and reference

formulations.

**14.1 Descriptive Statistics** 

Geometric mean, arithmetic mean, median, minimum, maximum, standard deviation and

coefficient of variation (arithmetic and geometric, respectively) will be calculated for each

PK parameter (C<sub>max</sub>, AUC<sub>0-t</sub> and T<sub>max</sub> for Paroxetine), logarithmically transformed and

untransformed.

For PK parameters C<sub>max</sub> and AUC<sub>0-t</sub> for Paroxetine, the following shall be calculated:

Difference of test and reference drugs.

• Quotient between test and reference drugs.

• The natural logarithm of the quotient between test and reference drugs.

• Histograms (ratios [A/B] and ln ratio [Ln (A/B)] will be performed.



Bioequivalence Pivotal Study Protocol of Paroxetine tablets 20 mg under fasting conditions.

# 14.2 Analysis of Variance

The In-transformed pharmacokinetic parameters (C<sub>max</sub>, AUC<sub>0-t</sub> for Paroxetine) will be analyzed using Type III sum of squares, with the main effects of formulation, period, sequence as fixed effects and subjects nested within sequence as a random effect. A separate ANOVA model will be used to analyze each of the parameters. The sequence effect will be tested at the 5% level of significance using the subjects nested within sequence mean square as the error term. Formulation and period effects will be tested at the 5% level of significance against the residual error (mean square error) from the ANOVA model as the error term. Each analysis of variance will include calculation of geometric least-squares means, the difference between the adjusted formulation means and the standard error associated with the difference.

#### 14.3 Statistical Model

The statistical model used in this research is a general linear model, whose equation is:

$$Y_{ijkl} = \mu + F_i + Seq_i + P_k + S_l (Seq_i) + e_{ijkl}$$

Where:

Y<sub>ijkl</sub> = Response of l<sup>th</sup> subject of j<sup>th</sup> Sequence when it received i<sup>th</sup> Formulation in k<sup>th</sup> Period

 $\mu$  = general mean

 $F_i$  = fixed effect of  $i^{th}$  formulation

 $Seq_i = fixed effect of i^{th} sequence$ 

 $P_k$  = fixed effect of  $k^{th}$  period

S<sub>1</sub> (Seq<sub>i</sub>)= random effect of l<sup>th</sup> subject nested within the i<sup>th</sup> sequence

 $e_{ijkl}$  = random error

# 14.4 Two One-Sided Test for Bioequivalence

A two one-sided test (Schuirmann) for the differences of least squares means between the formulations (test/reference) will be calculated for ln-transformed data of the C<sub>max</sub> and  $AUC_{0-t}$  for Paroxetine.

The hypothesis approach for the Schuirmann two one-sided test is:


Sponsor Code: 212969




Bioequivalence Pivotal Study Protocol of Paroxetine tablets 20 mg under fasting conditions.

Null hypothesis

 $H_0$ :  $\mu_{\text{test}} / \mu_{\text{ref}} < (0.8) H_{0a}$ :  $\mu_{\text{test}} / \mu_{\text{ref}} > (1.25)$  (not bioequivalent)

Alternative hypothesis  $H_1$ :  $\mu_{test} / \mu_{ref} \ge (0.8) H_{1a}$ :  $\mu_{test} / \mu_{ref} \le (1.25)$  (bioequivalent)

Acceptance criteria: to support bioequivalence, the null hypothesis in both conditions shall be rejected with a significance level of 5% for each side. With regards to the classical generated 90% confidence interval, it shall fall within the bioequivalence range of 80.00% -125.00%.

14.5 Statistical Power

Statistical power is the probability of rejecting the null hypothesis when it is false. Power is 1-Type II (where Type II error is the false negative error). The statistical power will be reported but considered only as informative when the test product is bioequivalent to the reference product.

14.6 Ratio Analysis

Ratio of geometric least squares means of the test and reference drugs will be computed for un-transformed and In-transformed primary pharmacokinetic parameters C<sub>max</sub> and AUC<sub>0-t</sub> for Paroxetine.

14.7 Intra-Subject Variability

Intra-subject variability will be computed for un-transformed data and for ln-transformed Pharmacokinetic parameters C<sub>max</sub> and AUC<sub>0-t</sub> for Paroxetine.

14.8 Analysis of Outliers

The outliers shall be identified (< -2.00 and > +2.00) using a  $\pm 2$  studentized residuals using the software SAS® version 9.4 or higher and their exclusion in the statistical analysis shall be justified (if applicable).

The subject's data will not be excluded from the statistical analysis exclusively due to mathematical or statistical reasons.

If statistical analysis concluded after removing the outliers, the results shall be submitted with and without the inclusion of outliers with a justification. In this case, the persons responsible




Bioequivalence Pivotal Study Protocol of Paroxetine tablets 20 mg under fasting conditions.

for the study, along with quality assurance personnel will investigate the possible causes of the appearance of outliers, and scientific evidence will be provided in addition to the statistical

evidence.

14.9 Criteria for elimination of subject data from the statistical analysis.

No data shall be eliminated from statistical analysis, except for the following.

a. Research (study) subjects with pre-dose concentrations in plasma:

If the pre-dose concentration is 5% of C<sub>max</sub> in that research subject, the data can be

included without adjustments in all pharmacokinetic measurements and calculations. In

cases where the pre-dose sample is >5% of the C<sub>max</sub>, the research subject shall be

eliminated from all bioequivalence assessments.

b. Data elimination due to vomiting or diarrhea.

Since the study drug is an immediate release product; the data from research subjects

who experience vomiting or diarrhea occur before 2 times the median t<sub>max</sub> or 2 times the

value of t<sub>max</sub> obtained in the research subject in a given period shall be eliminated from

all bioequivalence assessments.

c. A research subject who lacks measurable concentrations or with plasma concentrations

well below that of the reference drug.

A research subject is considered to have very low concentrations, if the AUC is less than

5% of the AUC geometric mean of the reference drug (shall be calculated without

inclusion of the atypical values of the research subject data). The exclusion of data due

to this reason will be accepted only with a scientific justification and with prior review

by COFEPRIS.

d. Since the planned study is a crossover and balanced, subjects who did not complete in

any of the study periods (subject that is discontinued or withdrawn) shall be eliminated

from all bioequivalence assessments.




Bioequivalence Pivotal Study Protocol of Paroxetine tablets 20 mg under fasting conditions.

The AUC<sub>0-t</sub> shall cover at least 80% of the AUC<sub>0-inf</sub>. The research subjects shall not be excluded

for the statistical analysis if the AUC<sub>0-t</sub> covers less than 80% of the AUC<sub>0-inf</sub>.

In case that a research subject elimination proceeds, according to the above-mentioned

information, the excluded research subject samples shall be analyzed and the results shall be

presented. Also, the statistical analysis shall be performed and shall be presented with and

without the data of eliminated research subjects.

14.10 Bioequivalence Criteria

Based on the statistical results of classic 90% confidence interval for the ratio of the geometric

least squares means for log-transformed PK parameters C<sub>max</sub> and AUC<sub>0-t</sub> for Paroxetine, a

conclusion will be drawn for test product (A) vs. the reference product (B) under fasting

conditions

The bioequivalence of the test product (A) with that of the reference product (B) under fasting

conditions will be concluded if the 90% confidence interval of the ratio of the test and

reference product (test/reference) falls within the acceptance range of 80.00 – 125.00% for

In-transformed PK parameters C<sub>max</sub> and AUC<sub>0-t</sub> of Paroxetine.

15.0 AMENDMENTS AND PROTOCOL DEVIATIONS

A protocol deviation is an unintended excursion from the approved protocol.

A major protocol deviation is a protocol deviation that may, as evaluated by the principal

investigator, or person designated by the investigator impact the safety of the subject or the

integrity of the trial. Major deviations will lead to withdrawal of a subject from the study...

Deviations not classified as major are considered as minor protocol deviations.

All protocol deviations should be reported to the sponsor by the Avant Santé and monitor (if

present on site) at the earliest possible time. The sponsor can propose to re-classify a protocol

deviation (minor to major or vice versa) upon evaluation. In such case, the classification made

by the sponsor prevails and will be communicated to Avant Santé together with a written

justification.

Sponsor Code: 212969




Bioequivalence Pivotal Study Protocol of Paroxetine tablets 20 mg under fasting conditions.

Major protocol deviations will only be implemented after sponsor's approval and obtaining approval or a favorable opinion from the Research Ethics Committee (REC) and Research

Committee (RC) and COFEPRIS.

The sponsor must be informed of minor protocol deviations, but before start of the following

clinical study period or before start of the bioanalytical phase/ statistical phase.

Minor protocol deviations will be reported sponsor and Committees if applicable, and will be

reported in study report:

• Logistic deviations (follow up visits that occurred outside the protocol required time

frame because of the participant's schedule etc.)

• All post dose in-house blood samples collected beyond  $\pm 2$  minutes during housing

period and  $\pm$  60 minutes for ambulatory samples from the scheduled collection time

will be reported as protocol deviations.

• Deviations related to meal consumption.

Administrative deviations (e.g. change of names).

Protocol deviation notification and reports are submitted to Health Authorities and/or relevant

Research Ethics Committee (REC) and Research Committee (RC) according to applicable

requirements/guidelines/law.

Procedure for documenting protocol deviations

The Principal Investigator, or person designated by PI, should document and explain any

deviation from the approved protocol. The notification of protocol deviation to sponsor can

be in exceptional cases communicated by verbal means (if immediate action/notification is

needed) and must be followed-up with written documentation (e.g. by e-mail; period update).

All major protocol deviations, as well as time point deviations or meal plan, must be described

in the final study report.


Sponsor Code: 212969




Bioequivalence Pivotal Study Protocol of Paroxetine tablets 20 mg under fasting conditions.

16.0 TERMINATION OF A STUDY

If the Principal Investigator terminates or suspends a study due to safety concerns,

investigator should inform the institution (Avant Santé) where applicable and the Principal

Investigator/institution should promptly inform the sponsor, subjects and the REC & RC.

If the sponsor terminates or suspends a study due to safety concerns to assure volunteers well-

being, the sponsor should promptly inform the institution/ Principal Investigator where

applicable and the investigator/institution should promptly inform the REC / RC and subjects.

If the REC / RC terminates or suspends its approval / favorable opinion of a trial / study, the

Principal Investigator should inform the institution where applicable and notify the sponsor.

The subjects would be informed on the reasons for the termination and compensated

adequately.

**Reasons for termination of study:** Principal Investigator / Sponsor / REC / RC / Sanitary

Responsible may discontinue / terminate the study at any time before study is complete. Some

of the reasons for these early terminations are:

1. A significant number of subjects are withdrawn from the study due to adverse events.

2. A significant number of subjects intermediately dropped out from the study / subjects

withdrew their consents to continue in the study, which may affect the overall power of

the study.

In case the sponsor finds that the investigational drug presents an unreasonable and significant

risk to subjects. In this case, the sponsor will discontinue the investigation as soon as possible,

and not later than 5 working days after making the decision. This will be communicated to

Principal Investigator, REC / RC and COFEPRIS.

17.0 DIRECT ACCESS TO SOURCE DATA/DOCUMENTS

The Quality Assurance (QA) personnel, Research Ethics Committee, Research Committee of

Avant Santé Research Center S.A. de C.V., sponsor/monitor and applicable regulatory




Bioequivalence Pivotal Study Protocol of Paroxetine tablets 20 mg under fasting conditions.

agencies (like Ministry of Health of México, COFEPRIS) will have access to the forms and

other source documents during inspection and audits.

**Source documents** 

Monitoring details describing strategy including definition of study critical data items and

processes, methods, responsibilities and requirements, including handling of noncompliance

issues and monitoring techniques (central, remote, or on-site monitoring) are provided in the

Monitoring Plan.

• Source documents provide evidence for the existence of the participant and substantiate the

integrity of the data collected. Source documents are filed at the investigator's site.

• Data reported on the CRF or entered in the eCRF that are transcribed from source documents

must be consistent with the source documents or the discrepancies must be explained. The

investigator may need to request previous medical records or transfer records, depending on

the study. Also, current medical records must be available.

Definition of what constitutes source data and its origin can be found in the Source Document

Acknowledgment.

• The investigator must maintain accurate documentation (source data) that supports the

information entered in the CRF.

• Study monitors will perform ongoing monitoring (remote or on-site) as per the Monitoring

Plan to confirm that data entered into the CRF by authorized site personnel are accurate,

complete, and verifiable from source documents; that the safety and rights of participants are

being protected; and that the study is being conducted in accordance with the currently

approved protocol and any other study agreements, ICH GCP, and all applicable regulatory

requirements.




Bioequivalence Pivotal Study Protocol of Paroxetine tablets 20 mg under fasting conditions.

18.0 QUALITY CONTROL AND QUALITY ASSURANCE

The raw data generated during the conduct of the study as well as the reports will undergo a

thorough Quality Control check and retrospective Quality Assurance audits performed by QA

personnel from Avant Santé Research Center, S.A. de C.V. to evaluate the conformity with

this protocol and all the governing SOPs.

The final report will contain a certification of the Quality Assurance Audit, duly signed by

the head of the Quality Assurance department.

19.0 INVESTIGATOR AND DELEGATION OF DUTIES

The Principal Investigator will ensure that the personnel involved in the study are adequately

qualified, trained and informed about the protocol, any amendment(s) made, the study drugs,

and their study-related duties and functions.

The investigator will maintain a list of the clinical investigator(s) and other appropriately

qualified personnel to whom he delegates significant study-related duties. The actual

delegation of the activities will be documented in the respective form and archived in the

RMF or trial master file.

20.0 ETHICAL CONSIDERATIONS

20.1 Ethical Standards

This study will be conducted in compliance with the requirements of NOM-177-SSA1-2013,

COFEPRIS guidelines, ICH-GCP and principles of Declaration of Helsinki (Fortaleza, Brazil,

October 2013).

Protocol, Case Report Form (CRF) and the informed consent form (ICF) approval will be

taken from the REC & RC, and COFEPRIS before initiation of the study.


Sponsor Code: 212969 Version No: 02 (12/Oct/2020)




Bioequivalence Pivotal Study Protocol of Paroxetine tablets 20 mg under fasting conditions.

20.2 Research Ethics Committee and Research Committee

This protocol, the informed consent form (ICF) and any other study-related material provided

to the subject will be reviewed and approved by REC & RC and the corresponding regulatory

agency.

The study will commence only after obtaining the written approval of the study protocol by

the REC/RC and COFEPRIS. Any modifications made to this protocol after its approval will

be presented to the REC/RC and COFEPRIS in accordance with the corresponding SOP and

any other regulatory requirement. A list of the changes in reference to the previous version

will be generated and included in the protocol as a "Change History" (Attachment-III).

**20.3 Informed Consent Process** 

The informed consent documents used during the informed consent process must be approved

by the REC / RC before providing to the subjects.

All subjects for this study will be provided a consent form describing this study and providing

sufficient information for subjects to make an informed decision about their participation in

this study. Extensive discussion of nature and objectives of the study, risks and possible

benefits of this study will be provided to each subject or subject's representative.

The designated study person will explain the details of the study to the subject or subject's

representative in a language that the subject or subject legal representative comprehends and

answer any questions that may arise. All volunteers shall sign the informed consent form

before their participation in the study. Each subject will be informed that they may withdraw

consent at any time throughout the course of the study.

A duplicate of the informed consent document will be given to the subjects. The subject has

the right to withdraw consent and discontinue further participation in the study. If the subject

decides to withdraw the study, subject will not face any penalties or loss of benefits to which

they may otherwise be entitled.




Bioequivalence Pivotal Study Protocol of Paroxetine tablets 20 mg under fasting conditions.

20.4 Subject Participation Compensation

The subjects will be compensated based on NOM 177-SSA1-2013 (COFEPRIS), and previous approval of REC/RC) on account of their participation in the study. In case of dropout / withdrawal of a subject because of a cause or decision of Avant Santé Research Center, S.A. de C.V. before study is concluded, the subjects will receive the full

compensation. In case the withdrawal is the result of any situation caused by the subject such

as non-compliance, discipline etc. compensation will be according to the conditions

established in the ICF, approved by the REC/RC.

20.5 Subject's Insurance

If a subject suffers any discomfort or injury, temporary or permanent, as a result of an event associated with the study drugs' administration, or that subject needs medical assistance, all the expenses will be met by the sponsor, through an insurance policy contracted by GlaxoSmithKline México, S.A. de C.V. Avant Santé Research Center S.A. de C.V. will ensure that if a subject needs emergency medical care, the same shall be provided at Tertiary care hospital, Swiss Hospital S.A.P.I. de C.V., contracted by Avant Santé Research Center

S.A. de C.V. If required, ambulance of Emergencia Médica Profesional, S. C. [contracted by

Avant Santé Research Center S.A. de C.V.] may be used for shifting the subject to Tertiary

care hospital.

If a subject suffers any discomfort or injury to medical practice will be covered by a valid civil liability insurance policy of Avant Santé Research Center S.A. de C.V. to the extent of

sum assured mentioned in the policy.

DATA HANDLING AND RECORD KEEPING 21.0

> All clinical data generated during the conduct of the study will be entered directly in the source documents as per the SOPs of Avant Santé Research Center S.A. de C.V. Raw data information will be transcribed in to electronic Case Report Form (eCRFs) according with SOP CP064 Source Data Management. All study (raw data and transcribed data) documents


Sponsor Code: 212969




Bioequivalence Pivotal Study Protocol of Paroxetine tablets 20 mg under fasting conditions.

will be reviewed for completeness by the PI or delegated personnel followed by QA personnel verification. The computer-generated data such as ECGs, randomization schedule, diagnostic lab reports will also be treated as raw data. All data related to the study will be in the custody of the PI until archived. All bioanalytical raw data generated and compiled by the study personnel during the conduct of the same will be reviewed for completeness. All data generated in the Bioanalytical Unit will be exported and transferred electronically based on C-DISC standards as recommended by GSK, to the Pharmacokinetics and Biostatistics

department for further evaluation.

21.1 Clinical Study Report

The Clinical study report will be prepared as per NOM-177-SSA1-2013 (COFEPRIS), Guía de Farmacovigilancia en Estudios clínicos, and sponsor requirements, having all the clinical,

bioanalytical, pharmacokinetic and statistical data subjected to Quality Assurance audits.

21.2 Confidentiality of Data

The data related to the subject identity will be kept confidential according to what it is described in the informed consent form and will be accessible only to the study personnel and if necessary, to the QA auditors, sponsor/monitors, REC/RC and COFEPRIS.

21.3 Archiving

The raw data and reports (this protocol, all data generated in connection to the study, along with a copy of this protocol, the signed ICFs, bioanalytical method validation report, concentration data, chromatograms and the final report) will be kept in the Trial Master Files together with all the records and documents pertaining to this study and they will be archived in the archives of Avant Santé Research Center S.A. de C.V. for at least 30 years based on GSK SOP POL-GSK-506-GRS GSK Global Records Retention Schedule - Version

7.

Avant Santé Research Center S.A. de C.V. will not destroy/discard any document related to the study without written confirmation from the sponsor.




Bioequivalence Pivotal Study Protocol of Paroxetine tablets 20 mg under fasting conditions.

21.4 Publication Policy

All data and results, and all intellectual property rights in data and results of the study will be

property of GlaxoSmithKline México, S.A. de C.V., who can use the same in different ways,

such as to be submitted to regulatory authorities or for being sent to other investigators.

The investigator, as long as he/she is free of using data from the study for scientific purposes,

shall discuss any publication with GlaxoSmithKline México, S.A. de C.V. prior to the same

and obtain the written consent from the sponsor regarding the publication.

This will be reviewed briefly and approval will not be delayed unnecessarily. In case of a

difference in opinion between sponsor and investigator(s), the content of publication will be

discussed with the objective of finding a solution that satisfies both parties

22.0 LIST OF ATTACHMENTS

Attachment-I: "Flowchart of Activities"

Attachment II: "Schedule of Events".

Sponsor Code: 212969

Attachment-III: "Change History".




Bioequivalence Pivotal Study Protocol of Paroxetine tablets 20 mg under fasting conditions.

#### 23.0 REFERENCES

- Summary of Product Characteristics (SmPC) of Paroxetine, film coated tablets 10 mg / 20 mg
   30 mg, last update in 13/09/2019, retrieved from https://www.medicines.org.uk/emc/product/7593
- 2. Drug information of Paxil (Paroxetine) 20 mg tablets, last updated on 01/04/2017, retrieved from
  - https://www.accessdata.fda.gov/drugsatfda docs/label/2017/020031s074lbl.pdf
- 3. "INFORME FARMACOCINÉTICO ESTADÍSTICO" of In-house study-AS/AO/ABR-17/0012 (Paroxetine 20 mg).
- 4. Bioequivalence Study of Paroxetine Hydrochloride Film-Coated Tablets; SHI Ai-ming, WANG Meng, ZHOU Wen-jia, ZHANG Quan-ying\*(Department of Pharmacy, The Second Affiliated Hospital of Soochow University, Suzhou 215004, China) and retrieved from; http://en.cnki.com.cn/Article en/CJFDTOTAL-ZGYX201205014.htm
- 5. Oficio Circular CAS/OR/01/868/2013 "Lineamientos por los que se establecen los requisitos para cambio de fabricante de fármaco o inclusión de fabricantes en México.
- 6. NORMA Oficial Mexicana NOM-059-SSA1-2015, Buenas prácticas de fabricación de medicamentos. 30/Jun/2015.
- 7. NORMA Oficial Mexicana NOM-177-SSA1-2013, Que establece las pruebas y procedimientos para demostrar que un medicamento es intercambiable. Requisitos a que deben sujetarse los Terceros Autorizados que realicen las pruebas de intercambiabilidad. Requisitos para realizar los estudios de biocomparabilidad. Requisitos a que deben sujetarse los Terceros Autorizados, Centros de Investigación o Instituciones Hospitalarias que realicen las pruebas de biocomparabilidad, Sep, 2013.
- 8. Guideline for Good Clinical Practice, E6 (R2), International Council on Harmonization of Technical Requirements for Registration of Pharmaceuticals for Human use, Current Step 4 version, 09 November 2016.


Sponsor Code: 212969




#### Bioequivalence Pivotal Study Protocol of Paroxetine tablets 20 mg under fasting conditions.

- 9. NORMA Oficial Mexicana NOM-220-SSA1-2016, Instalación y operación de la farmacovigilancia, 19/07/2017 y modificaciones a la NOM-220-SSA1-2016 con fecha de 30/09/2020.
- 10. Reglamento de la Ley General de Salud en Materia de Investigación, Feb, 1984.
- 11. NORMA Oficial Mexicana NOM-012-SSA3-2012, Que establece los criterios para la ejecución de proyectos de investigación para la salud en seres humanos, 04/01/2013.
- 12. "Guía de Farmacovigilancia en Investigación clínica", vigente
- 13. (Guía para Bioequivalencia) "Guía para sometimiento de protocolos de investigación para demostrar la intercambiabilidad de medicamentos" obtenido de http://www.cofepris.gob.mx/AS/Paginas/Mol%C3%A9culas%20nuevas/Tr%C3%A1mites-PI.aspx
- 14. EMEA-GUIDELINE ON THE INVESTIGATION OF BIOEQUIVALENCE- London, 20 January 2010.
- 15. Food and Drug Administration (FDA), Guidance for Industry: Statistical approaches to establishing bioequivalence 2001.
- 16.Guidance on Study Design Considerations Related to COVID-19 for new GSK Clinical Trials v1 26May20


Sponsor Code: 212969


CONFIDENTIAL Avant Santé Research Center S.A. de C.V



#### Bioequivalence Pivotal Study Protocol of Paroxetine tablets 20 mg under fasting conditions.




> CONFIDENTIAL Avant Santé Research Center S.A. de C.V



Bioequivalence Pivotal Study Protocol of Paroxetine tablets 20 mg under fasting conditions.

# **ATTACHMENT-II**

# **SCHEDULE OF EVENTS**

# **SCREENING**

| Day | Hours | Scheduled Time | Activity |
|---|---|---|---|
| | | | Informed consent for screening and/or study. |
| -90 | | | Recording of weight and height. |
| days<br>to<br>day - | N/A | N/A | Medical and Physical examination. Subject's well-being assessment. |
| | | | Laboratory: hematology, blood chemistry, urinalysis; serology; alcohol testing, urine test for drugs; pregnancy test in urine: ECG. |
| 1 | | | Evaluation of inclusion and exclusion criteria. |
| -72 h | N/A | N/A | RT-PCR test for the detection and diagnosis of SARS-COV-2 |

# **PERIOD 1**

| Day | Hours | Scheduled Time* | Activity |
|---|---|---|---|
| | -20.0010.50 | 12:00 – 21:30 | Arrival in clinical facilities. Evaluation of inclusion and exclusion criteria based on screening tests (demography, medical history, physical examination findings, ECG, laboratory tests and RT-PCR). |
| -1 | | | Breath alcohol testing, urine drug screen, urine pregnancy test for females, medical & physical examination, vital signs recording, prior and concomitant medication and well-being assessment and admission into clinics (Check-in). |
| | -10.50 to -10.00 | 21:30-22:00 | Dinner. |
| | -3.00 | 05:00 | Wakeup time, bath following by pre-dose Medical examination, Vital signs recording and well-being assessment. |
| | -1.50 to 0.00 | 06:30 - 08:00 | Cannulation and 1st blood sample (pre-dose 0.00 h) collection |
| | - 1.00 to 2.00 | 07:00 to 10:00 | Water restriction period. |
| | 0.00 | 08:00 | Dosing (administration of test or reference product) with 250 mL of water. |
| 1 | 0.00 to 2.00 | 08:00 to 10:00 | Posture restriction period. |
| 1 | 00.50 | 08:30 | 2 <sup>nd</sup> blood sample collection. |
| | 01.00 | 09:00 | 3 <sup>rd</sup> blood sample collection. |
| | 01.50 | 09:30 | 4 <sup>th</sup> blood sample collection |
| | 02.00 | 10:00 | 5 <sup>th</sup> blood sample collection, |
| | 02.50 | 10:30 | 6 <sup>th</sup> blood sample collection. |
| | 03.00 | 11:00 | 7 <sup>th</sup> blood sample collection, Vital signs recording and well-being assessment. |




Sponsor Code: 212969

Format No.: CPF127-03E No. Reference SOP: CP006

# Bioequivalence Pivotal Study Protocol of Paroxetine tablets 20 mg under fasting conditions.

| Day | Hours | Scheduled Time* | Activity |
|---|---|---|---|
| | 03.50 | 11:30 | 8 <sup>th</sup> blood sample collection. |
| | 04.00 | 12:00 | 9 <sup>th</sup> blood sample collection. Lunch. |
| | 04.50 | 12:30 | 10 <sup>th</sup> blood sample collection. |
| | 05.00 | 13:00 | 11 <sup>th</sup> blood sample collection, Vital signs recording and well-being assessment. |
| | 05.50 | 13:30 | 12 <sup>th</sup> blood sample collection. |
| | 06.00 | 14:00 | 13 <sup>th</sup> blood sample collection. |
| | 06.50 | 14:30 | 14 <sup>th</sup> blood sample collection |
| | 07.00 | 15:00 | 15 <sup>th</sup> blood sample collection. |
| | 08.00 | 16:00 | 16 <sup>th</sup> blood sample collection, Snacks. |
| | 09.00 | 17:00 | 17 <sup>th</sup> blood sample collection. |
| | 10.00 | 18:00 | 18 <sup>th</sup> blood sample collection. |
| | 12.00 | 20:00 | 19 <sup>th</sup> blood sample collection, Vital signs recording and well-being assessment, Dinner. |
| | 16.00 | 00:00 | 20 <sup>th</sup> blood sample collection. |
| 2 | 24.00 | 08:00 | 21 <sup>th</sup> blood sample collection. Medical examination with vital signs, well-being assessment and exit from clinics (Check-out). |
| | 36.00 | 20:00 | 22 <sup>nd</sup> blood sample collection, well-being assessment and vital signs recording. |
| 3 | 48.00 | 08:00 | 23 <sup>nd</sup> blood sample collection, well-being assessment and vital signs recording. |
| 4 | 72.00 | 08:00 | 24 <sup>nd</sup> blood sample collection, well-being assessment and vital signs recording. |

<sup>\*</sup>The schedule of events may change according to the dosing time <sup>a:</sup> Update of changes since screening visit

| Washout | There will be a washout period of at least 7 days between successive dosing. Subjects will be instructed to self-quarantine during the outpatient period of the |
|---|---|
| Period | study and to monitor at home their daily body temperature |

#### PERIOD 2

| Day | Hours | Scheduled Time* | Activity |
|---|---|---|---|
| | | | Arrival in clinical facilities. |
| -1 | -20.0010.50 | 12:00 – 21:30 | Breath alcohol testing, urine drug screen, urine pregnancy test for females, medical & physical examination, vital signs recording, prior and concomitant medication and well-being assessment and admission into clinics (Check-in). |
| | -10.50 to -10.00 | 21:30-22:00 | Dinner. |


> CONFIDENTIAL Avant Santé Research Center S.A. de C.V



#### Bioequivalence Pivotal Study Protocol of Paroxetine tablets 20 mg under fasting conditions.

| Day | Hours | Scheduled Time* | Activity |
|---|---|---|---|
| | -3.00 | 05:00 | Wakeup time, bath following by pre-dose Medical examination, Vital signs recording and well-being assessment. |
| | -1.50 to 0.00 | 06:30 - 08:00 | Cannulation and 1 <sup>st</sup> blood sample (pre-dose 0.00 h) collection |
| | - 1.00 to 2.00 | 07:00 to 10:00 | Water restriction period. |
| | 0.00 | 08:00 | Dosing (administration of test or reference product) with 250 mL of water. |
| | 0.00 to 2.00 | 08:00 to 10:00 | Posture restriction period. |
| | 00.50 | 08:30 | 2 <sup>nd</sup> blood sample collection. |
| | 01.00 | 09:00 | 3 <sup>rd</sup> blood sample collection. |
| | 01.50 | 09:30 | 4 <sup>th</sup> blood sample collection |
| | 02.00 | 10:00 | 5 <sup>th</sup> blood sample collection, |
| | 02.50 | 10:30 | 6 <sup>th</sup> blood sample collection. |
| | 03.00 | 11:00 | 7 <sup>th</sup> blood sample collection, Vital signs recording and well-being assessment. |
| 1 | 03.50 | 11:30 | 8 <sup>th</sup> blood sample collection. |
| | 04.00 | 12:00 | 9 <sup>th</sup> blood sample collection. Lunch. |
| | 04.50 | 12:30 | 10 <sup>th</sup> blood sample collection. |
| | 05.00 | 13:00 | 11th blood sample collection, Vital signs recording and well-being assessment. |
| | 05.50 | 13:30 | 12 <sup>th</sup> blood sample collection. |
| | 06.00 | 14:00 | 13 <sup>th</sup> blood sample collection. |
| | 06.50 | 14:30 | 14 <sup>th</sup> blood sample collection |
| | 07.00 | 15:00 | 15 <sup>th</sup> blood sample collection. |
| | 08.00 | 16:00 | 16 <sup>th</sup> blood sample collection, Snacks. |
| | 09.00 | 17:00 | 17 <sup>th</sup> blood sample collection. |
| | 10.00 | 18:00 | 18 <sup>th</sup> blood sample collection. |
| | 12.00 | 20:00 | 19 <sup>th</sup> blood sample collection, Vital signs recording and well-being assessment, Dinner. |
| | 16.00 | 00:00 | 20 <sup>th</sup> blood sample collection. |
| 2 | 24.00 | 08:00 | 21 <sup>th</sup> blood sample collection. Medical examination with vital signs, well-being assessment and exit from clinics (Check-out). |
| | 36.00 | 20:00 | 22 <sup>nd</sup> blood sample collection, well-being assessment and vital signs recording. |
| 3 | 48.00 | 08:00 | 23 <sup>nd</sup> blood sample collection, well-being assessment and vital signs recording. |
| 4 | 72.00 | 08:00 | 24 <sup>nd</sup> blood sample collection, well-being assessment and vital signs recording. Final Compensation for subjects (applicable only for period 2). |

Seven (7) to 9 days after the collection of 72-h blood sample in second period or after the withdrawal, a telephone call will be made to each subject by the personnel designated by the PI to monitor any serious adverse event, specifically, subjects will be questioned about any symptoms related to COVID-19.

Sponsor Code: 212969


<sup>\*</sup>The schedule of events may change according to the dosing time



Bioequivalence Pivotal Study Protocol of Paroxetine tablets 20 mg under fasting conditions.

# ATTACHMENT-III CHANGE HISTORY

| Current | Supersedes, | Changes Made |
|---|---|---|
| Version No. | Effective Date | Changes Made |
| 01 | N/A | N/A |
| 02 | 01,<br>10/Jan/2020 | 1. Format number "CPF127-02E" of the protocol is modified to "CPF127-03E" 2. The Sanitary Responsible of Clinical Unit is modified on page 6. 3. COVID-19, SARS-CoV-2 and RT-PCR are added to abbreviations. 4. The address of the Clinical Diagnostic Laboratory is modified in section 2.3. 5. Real-time (RT-PCR) test for the detection and diagnosis of SARS-COV-2 is added in section 1.0 and 8.1 Screening (selection and enrollment). 6. "Have a negative test for active COVID-19, within 72 hours prior to the first period check-in. The testing should be done using a molecular (RT-PCR) approved by the country regulatory authorities" is added in section 8.3 (Inclusion criteria). 7. "Subjects with symptoms suggestive of active COVID-19 infection (i.e. fever, cough, respiratory difficulties) within 14 days of inpatient admission" and "Subjects with known COVID-19 positive contacts* within the past 14 days prior to the first period check-in. *Positive Contact; this means, if the subject has |


Sponsor Code: 212969


CONFIDENTIAL Avant Santé Research Center S.A. de C.V



#### Bioequivalence Pivotal Study Protocol of Paroxetine tablets 20 mg under fasting conditions.

- been living, providing, care, being within 1.5 m for at least 15 min or having exposure to respiratory secretions with/to a person who has COVID-19" is added in section 8.3 (Exclusion criteria).
- 8. In section 8.5, criteria b is added "In case a subject is positive for COVID-19 or has a related symptom (i.e. fever, cough, respiratory difficulties), they shall be isolated for 14 days and they shall be discontinued In case any other subject was exposed to a COVID-19 patient, they must report this to Avant Santé, GSK and/or their primary care provider".
- 9. In section 9.3 is added "Recommendations during washout period and visits to the center (ambulatory samples)".
- 10. "Subjects will be instructed to self-quarantine during the outpatient period of the study i.e. until 72 h blood sample collection in period-2 or until withdrawal, whichever is earlier, and to monitor at home their daily body temperature" is added in section 1.0 and 9.4 (Housing).
- 11. The assessment of vital signs at the time of ambulatory samples is added in section 1.0 and 11.1 (Assessment of safety).
- 12. "Seven (7) to 9 days after the collection of 72-h sample in second period or after withdrawal, a telephone call will be made to each subject by the personnel




#### Bioequivalence Pivotal Study Protocol of Paroxetine tablets 20 mg under fasting conditions.

- designated by the PI to monitor any adverse event, specifically, subjects will be questioned about any symptoms related to COVID-19" is added in section 1.0 and 11.1 (Assessment of safety).
- 13. The period of recording AEs "(i.e., within 7 or 9 days after the last sample collection or after withdrawal)" is added in section 11.2 (Recording of AEs).
- 14. The section 11.2 "The notification through the platform assigned by the CNFV for this purpose shall be performed as soon as possible but no more than 7 calendar days \* from the time of awareness" is modified by "The notification through the platform assigned by the CNFV for this purpose shall be performed according to the timelines stablished in the valid NOM-220-SSA1-2016".
- 15. Typo errors are corrected in section 14.4.
- 16. Information regarding "source documents" was added in section 17.0.
- 17. In section 20.3 "a copy of the informed consent ..." is modified by "a duplicate of the informed consent ..."
- 18. Reference 9 is updated and reference 16 is added.
- 19. Attachment-I (Flowchart of activities) is updated.
- 20. Attachment-II (Schedule of events) is updated based on the new information provided above.


Various No. 02 (12/Oct/2020)


Sponsor Code: 212969

